CLINICAL TRIAL: NCT03525678
Title: A Phase II, Open Label, Randomized, Two-Arm Study to Investigate the Efficacy and Safety of Two Doses of the Antibody Drug Conjugate GSK2857916 in Participants With Multiple Myeloma Who Had 3 or More Prior Lines of Treatment, Are Refractory to a Proteasome Inhibitor and an Immunomodulatory Agent and Have Failed an Anti-CD38 Antibody (DREAMM 2)
Brief Title: A Study to Investigate the Efficacy and Safety of Two Doses of GSK2857916 in Participants With Multiple Myeloma Who Have Failed Prior Treatment With an Anti-CD38 Antibody
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205678; 2017-004810-25 (EudraCT Number)
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Results first posted 2020-04-28 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: Relapsed Refractory multiple myeloma; Antibody-drug conjugate; Patient-Reported Outcome Version of the Common Term Criteria for Adverse Events; Quality of Life Questionnaire 20-item Multiple Myeloma module; Multiple Myeloma; Quality of Life Questionnaire 30-item Core module
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Participants receiving frozen 2.5 mg/kg belantamab mafodotin (Experimental): Participants will receive 2.5 mg/kg frozen liquid belantamab mafodotin. Participants will be administered with frozen liquid belantamab mafodotin via infusion pump every 3 weeks.
  Interventions: Drug: Belantamab mafodotin frozen liquid
- Participants receiving frozen 3.4 mg/kg belantamab mafodotin (Experimental): Participants will receive 3.4 mg/kg frozen liquid belantamab mafodotin. Participants will be administered with frozen liquid belantamab mafodotin via infusion pump every 3 weeks.
  Interventions: Drug: Belantamab mafodotin frozen liquid
- Participants receiving lyophilized belantamab mafodotin (Experimental): Participants in lyophilized arm will receive lyophilized belantamab mafodotin once lyophilized configuration becomes available and enrollment has been completed for frozen liquid arms.
  Interventions: Drug: Belantamab mafodotin lyophilized powder

INTERVENTIONS:
Drug: Belantamab mafodotin frozen liquid — Belantamab mafodotin will be available as frozen liquid. Frozen liquid will be available as 30 milligram (mg)/vial solution in a single use vial with unit dose strength of 2.5 or 3.4 mg/kg. Belantamab mafodotin will be administered as IV solution over at least 30 minutes. Frozen belantamab mafodotin will be diluted in 0.9 percent saline and administered via infusion pump.
  Arms: Participants receiving frozen 2.5 mg/kg belantamab mafodotin; Participants receiving frozen 3.4 mg/kg belantamab mafodotin
Drug: Belantamab mafodotin lyophilized powder — Belantamab mafodotin will be available as lyophilized powder. Lyophilized powder will be available as 100 mg/vial in single-use vial for reconstitution with unit dose strength of 3.4 mg/kg. Lyophilized belantamab mafodotin will be reconstituted using water for injection and diluted with saline before use.
  Arms: Participants receiving lyophilized belantamab mafodotin

SUMMARY:
Multiple myeloma (MM) is an incurable malignancy and accounts for 1 percentage (%) of all cancers and for 10% of all hematologic malignancies. Participants with relapsed/refractory multiple myeloma (RRMM) will be included in this study, to evaluate the efficacy and safety of belantamab mafodotin (GSK2857916) monotherapy. Participants will be treated with belantamab mafodotin monotherapy until disease progression (PD) or unacceptable toxicity and will be followed for Progression Free Survival and Overall survival. The participants will be randomized to receive either frozen belantamab mafodotin at the dose of 2.5 milligram per kilogram (mg/kg) or 3.4 mg/kg administered Intravenously (IV). There will be an independent cohort of participants who will receive a lyophilized configuration of belantamab mafodotin. For participants who discontinued from the study other than Progressive disease (PD), disease evaluation will continue to be performed at 3-week intervals until confirmed PD, death, start of a new anticancer treatment, withdrawal of consent, or end of the study whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Participants who provided signed written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Male or female, 18 years or older.
* Participants with Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Participants with histologically or cytologically confirmed diagnosis of MM as defined in IMWG, 2014 criteria, and participant has undergone stem cell transplant or is considered transplant ineligible and has failed at least 3 prior lines of anti-myeloma treatments, including an anti-CD38 antibody (example [e.g.], daratumumab) alone or in combination, and is refractory to an Immunomodulatory drug (IMiD) (that is [i.e.], lenalidomide or pomalidomide), and to a proteasome inhibitor (e.g., bortezomib, ixazomib or carfilzomib).
* The participant has measurable disease with at least one of the following: Serum M-protein >=0.5 grams per deciliter (g/dL) (>=5 grams per Liter [g/L]); Urine M-protein >=200 milligram per 24 hours (mg/24h); Serum Free light chain (FLC) assay: Involved FLC level >=10 mg/dL (>=100 mg/Liter) and an abnormal serum FLC ratio (<0.26 or >1.65).
* Participants with a history of autologous stem cell transplant are eligible for study participation provided the following eligibility criteria are met: transplant was >100 days prior to study enrollment; no active infection(s); participants meet the remainder of the eligibility criteria outlined in the protocol.
* Participants with adequate organ system functions as defined follows: Absolute neutrophil count (ANC) >=1.0 X 10^9/L; Hemoglobin >=8.0 g/dL; Platelets>= 50 X 10^9/L; Total bilirubin <=1.5X Upper limit of normal (ULN). Isolated bilirubin >=1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent); Alanine aminotransferase (ALT) <=2.5X ULN; Estimated glomerular filtration rate (eGFR) >=30 milliliter per minute per 1.73 meter square (mL/min/m^2); Spot urine (albumin/creatinine ratios [spot urine]) <500 milligram per gram (mg/g) (56 mg per millimoles [mg/mmol]); Left ventricular ejection fraction (LVEF) (Echocardiogram)>=45 percent.
* Female participants: Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breastfeeding, and not a woman of childbearing potential (WOCBP) or is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency, during the intervention period and for at least 80 days after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. A WOCBP must have a negative highly sensitive serum pregnancy test (as required by local regulations) within 72 hours before the first dose of study intervention. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Male participants: Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Male participants are eligible to participate if they agree to the following during the intervention period and for at least 140 days: Refrain from donating sperm; Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent; or Agree to use a male condom and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year as when having sexual intercourse with a WOCBP who is not currently pregnant.
* All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events [NCI-CTCAE]), version 4.03, must be <=Grade 1 at the time of enrollment except for alopecia and Grade 2 peripheral neuropathy.
* For France only: A participant will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Systemic anti-myeloma therapy within <=14 days, or 5 half-lives, whichever is shorter, or plasmapheresis within 7 days prior to the first dose of study drug.
* Systemic treatment with high dose steroids (equivalent to >=60 mg prednisone daily for >=4 days) within the past 14 days if administered to treat MM or non-MM disease.
* Symptomatic amyloidosis, active 'polyneuropathy, organomegaly, endocrinopathy, myeloma protein, and skin changes' (POEMS) syndrome, active plasma cell leukemia at the time of screening.
* Prior allogeneic stem cell transplant.
* Current corneal epithelial disease except mild punctate keratopathy.
* Use of an investigational drug within 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug. Prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drugs. Prior B-cell maturation antigen (BCMA) targeted therapy.
* Evidence of active mucosal or internal bleeding.
* Any major surgery within the last four weeks.
* Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM are eligible.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Malignancies other than disease under study are excluded, except for any other malignancy from which the participant has been disease-free for more than 2 years and, in the opinion of the principal investigators and GlaxoSmithKline Medical Monitor, will not affect the evaluation of the effects of this clinical trial treatment on the currently targeted malignancy (MM). Participants with curatively treated non-melanoma skin cancer may be enrolled.
* Evidence of cardiovascular risk including any of the following: Corrected QT interval Fridericia (QTcF) interval >480 milliseconds (msec); Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant electrocardiogram abnormalities such as 2nd degree (Type II) or 3rd degree atrioventricular (AV) block; History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within six months of Screening; Class III or IV heart failure as defined by the New York Heart Association functional classification system (NYHA); Uncontrolled hypertension.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
* Pregnant or lactating female.
* Active infection requiring antibiotic, antiviral, or antifungal treatment.
* Known Human Immunodeficiency Virus (HIV) infection.
* Presence of hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb at screening or within 3 months prior to first dose of study treatment.
* Positive hepatitis C antibody test result or positive hepatitis C Ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2024-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (55):
- United States (18):
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Fairway, Kansas
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Madison, Wisconsin
- Australia (3):
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Melbourne, Victoria
- Canada (3):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Toronto, Ontario
- France (6):
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Toulouse
- Germany (6):
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, Koblenz
  - GSK Investigational Site, Schwerin
  - GSK Investigational Site, Tübingen
  - GSK Investigational Site, Würzburg
- Italy (4):
  - GSK Investigational Site, Aviano PN
  - GSK Investigational Site, Parma
  - GSK Investigational Site, Rionero in Vulture PZ
  - GSK Investigational Site, Torino
- Spain (8):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, PamplonaNavarra
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Valencia
- United Kingdom (7):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bournemouth
  - GSK Investigational Site, London
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Stoke-on-Trent
  - GSK Investigational Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Lonial S, Lee HC, Badros A, Trudel S, Nooka AK, Chari A, Abdallah AO, Callander N, Lendvai N, Sborov D, Suvannasankha A, Weisel K, Karlin L, Libby E, Arnulf B, Facon T, Hulin C, Kortum KM, Rodriguez-Otero P, Usmani SZ, Hari P, Baz R, Quach H, Moreau P, Voorhees PM, Gupta I, Hoos A, Zhi E, Baron J, Piontek T, Lewis E, Jewell RC, Dettman EJ, Popat R, Esposti SD, Opalinska J, Richardson P, Cohen AD. Belantamab mafodotin for relapsed or refractory multiple myeloma (DREAMM-2): a two-arm, randomised, open-label, phase 2 study. Lancet Oncol. 2020 Feb;21(2):207-221. doi: 10.1016/S1470-2045(19)30788-0. Epub 2019 Dec 16. PMID 31859245
- [Background] Prawitz T, Popat R, Suvannasankha A, Sarri G, Hughes R, Wang F, Hogea C, Ferrante SA, Gorsh B, Willson J, Kapetanakis V. DREAMM-2: Indirect Comparisons of Belantamab Mafodotin vs. Selinexor + Dexamethasone and Standard of Care Treatments in Relapsed/Refractory Multiple Myeloma. Adv Ther. 2021 Nov;38(11):5501-5518. doi: 10.1007/s12325-021-01884-7. Epub 2021 Sep 24. PMID 34561812
- [Background] Nooka AK, Cohen AD, Lee HC, Badros A, Suvannasankha A, Callander N, Abdallah AO, Trudel S, Chari A, Libby EN, Chaudhry M, Hultcrantz M, Kortum KM, Popat R, Sborov D, Hakim S, Lewis E, Gorsh B, Bhushan B, McKeown A, Gupta I, Opalinska J, Richardson PG, Lonial S. Single-agent belantamab mafodotin in patients with relapsed/refractory multiple myeloma: Final analysis of the DREAMM-2 trial. Cancer. 2023 Dec 1;129(23):3746-3760. doi: 10.1002/cncr.34987. Epub 2023 Aug 25. PMID 37622738
- [Derived] Collins J, van Noort M, Rathi C, Post TM, Struemper H, Jewell RC, Ferron-Brady G. Longitudinal efficacy and safety modeling and simulation framework to aid dose selection of belantamab mafodotin for patients with multiple myeloma. CPT Pharmacometrics Syst Pharmacol. 2023 Oct;12(10):1411-1424. doi: 10.1002/psp4.13016. Epub 2023 Aug 2. PMID 37465991
- [Derived] Nikolaou A, Ambavane A, Shah A, Ma W, Tosh J, Kapetanakis V, Willson J, Wang F, Hogea C, Gorsh B, Gutierrez B, Sapra S, Suvannasankha A, Samyshkin Y. Belantamab mafodotin for the treatment of relapsed/refractory multiple myeloma in heavily pretreated patients: a US cost-effectiveness analysis. Expert Rev Hematol. 2021 Dec;14(12):1137-1145. doi: 10.1080/17474086.2021.1970522. Epub 2021 Sep 20. PMID 34465265
- [Derived] Lonial S, Lee HC, Badros A, Trudel S, Nooka AK, Chari A, Abdallah AO, Callander N, Sborov D, Suvannasankha A, Weisel K, Voorhees PM, Womersley L, Baron J, Piontek T, Lewis E, Opalinska J, Gupta I, Cohen AD. Longer term outcomes with single-agent belantamab mafodotin in patients with relapsed or refractory multiple myeloma: 13-month follow-up from the pivotal DREAMM-2 study. Cancer. 2021 Nov 15;127(22):4198-4212. doi: 10.1002/cncr.33809. Epub 2021 Jul 27. PMID 34314018
- [Derived] Lonial S, Nooka AK, Thulasi P, Badros AZ, Jeng BH, Callander NS, Potter HA, Sborov D, Zaugg BE, Popat R, Degli Esposti S, Byrne J, Opalinska J, Baron J, Piontek T, Gupta I, Dana R, Farooq AV, Colby K, Jakubowiak A. Management of belantamab mafodotin-associated corneal events in patients with relapsed or refractory multiple myeloma (RRMM). Blood Cancer J. 2021 May 26;11(5):103. doi: 10.1038/s41408-021-00494-4. PMID 34039952
- [Derived] Farooq AV, Degli Esposti S, Popat R, Thulasi P, Lonial S, Nooka AK, Jakubowiak A, Sborov D, Zaugg BE, Badros AZ, Jeng BH, Callander NS, Opalinska J, Baron J, Piontek T, Byrne J, Gupta I, Colby K. Corneal Epithelial Findings in Patients with Multiple Myeloma Treated with Antibody-Drug Conjugate Belantamab Mafodotin in the Pivotal, Randomized, DREAMM-2 Study. Ophthalmol Ther. 2020 Dec;9(4):889-911. doi: 10.1007/s40123-020-00280-8. Epub 2020 Jul 25. PMID 32712806

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, randomized, multicenter study to evaluate the efficacy and safety of belantamab mafodotin monotherapy at a dose of 2.5 milligram per kilogram (mg/kg) or 3.4 mg/kg, given intravenously (IV) in participants with relapsed/refractory multiple myeloma (RRMM).
Pre-assignment Details: A total of 221 participants were enrolled in this study. The study consisted of two phases - Main Study Phase and Post Analysis Continued Treatment (PACT) Phase. In PACT phase those participants benefiting from drug continued to receive study drug until discontinuation or withdrawal from study.
Groups:
- Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid): Participants were administered frozen liquid (30 mg/vial solution in a single use vial) at a dose of 2.5 mg/kg GSK2857916 as IV solution once every three weeks for a maximum of up to 39 cycles (1 cycle= 21 days). Frozen liquid was diluted with 0.9 percent saline.
- Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid): Participants were administered frozen liquid (30 mg/vial solution in a single use vial) at a dose of 3.4 mg/kg GSK2857916 as IV solution once every three weeks for a maximum of up to 32 cycles (1 cycle= 21 days). Frozen liquid was diluted with 0.9 percent saline.
- Main Study: GSK2857916 3.4 mg/kg (Lyophilized): Participants were administered lyophilized powder (100 mg/vial in a single use vial) at a dose of 3.4 mg/kg GSK2857916 given IV for a maximum of 35 cycles (1 cycle= 21 days). Lyophilized powder was reconstituted using water for injection.
- PACT Phase: GSK2857916 2.5 mg/kg (Frozen Liquid): Participants were administered frozen liquid (30 mg/vial solution in a single use vial) at a dose of 2.5 mg/kg GSK2857916 as IV solution once every three weeks up to approximately 101 weeks. Frozen liquid was diluted with 0.9 percent saline.
- PACT Phase: GSK2857916 3.4 mg/kg (Frozen Liquid): Participants were administered frozen liquid (30 mg/vial solution in a single use vial) at a dose of 3.4 mg/kg GSK2857916 as IV solution once every three weeks up to approximately 101 weeks. Frozen liquid was diluted with 0.9 percent saline.
Period: Main Study (Day 1 to 186 Weeks)
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized) | PACT Phase: GSK2857916 2.5 mg/kg (Frozen Liquid) | PACT Phase: GSK2857916 3.4 mg/kg (Frozen Liquid)
Started | 97 | 99 | 25 | 0 | 0
Received Study Treatment | 95 | 99 | 24 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 97 | 99 | 25 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 2 | 2 | 0 | 0
Not completed — Physician Decision | 2 | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 2 | 0 | 0
Not completed — Death | 70 | 80 | 16 | 0 | 0
Not completed — other reasons | 14 | 10 | 5 | 0 | 0
Not completed — Transitioned to PACT phase | 1 | 2 | 0 | 0 | 0
Period: PACT Phase (From 186 Weeks to 325 Weeks)
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized) | PACT Phase: GSK2857916 2.5 mg/kg (Frozen Liquid) | PACT Phase: GSK2857916 3.4 mg/kg (Frozen Liquid)
Started | 0 | 0 | 0 | 1 (Participant transitioned from main study phase to PACT Phase.) | 2 (Participants transitioned from main study phase to PACT Phase.)
Completed | 0 | 0 | 0 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were presented for all randomized participants including 3 randomized participants who never received treatment (2-withdrawal by physician decision and 1-death).
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized) | Total
Number analyzed (Participants) | 97 | 99 | 25 | 221
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (10.01) | 66.0 (9.09) | 67.2 (10.78) | 65.3 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 43 | 11 | 100
  Male | 51 | 56 | 14 | 121
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 16 | 11 | 3 | 30
  Asian - Central/South Asian Heritage | 1 | 0 | 0 | 1
  Asian - East Asian Heritage | 1 | 0 | 0 | 1
  Asian - South East Asian Heritage | 0 | 1 | 1 | 2
  White - Arabic/North African Heritage | 4 | 2 | 0 | 6
  White - White/Caucasian/European Heritage | 72 | 83 | 21 | 176
  Mixed Asian Race | 0 | 1 | 0 | 1
  Mixed White Race | 0 | 1 | 0 | 1
  Unknown | 1 | 0 | 0 | 1
  Missing | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) by Independent Review Committee (IRC) (Full Analysis Population)
Description: ORR was determined according to the 2016 international myeloma working group (IMWG) response criteria by IRC. ORR was calculated as the percentage of participants with a confirmed partial response (PR) or better (that is [i.e.], PR, very good partial response [VGPR], complete response [CR] and stringent complete response [sCR]). Confidence intervals were based on the exact method.
Time Frame: Up to 48 weeks
Population: Full Analysis Population comprised of all randomized participants (any participant who received a treatment randomization number was considered as randomized) whether or not randomized treatment was administered. This population was based on the treatment the participant was randomized to.
Measure: Number (97.5% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 97 | 99 | 25
Percentage of Participants | 31 [20.8 to 42.6] | 34 [23.9 to 46.0] | 48 [25.5 to 71.1]

2. Primary Outcome: Overall Response Rate by Independent Review Committee (Efficacy Population)
Description: ORR was determined according to the 2016 IMWG response criteria by IRC. ORR was calculated as the percentage of participants with a confirmed PR or better (i.e., PR, VGPR, CR and sCR). Confidence intervals were based on the exact method. Efficacy Population comprised of first 130 intent-to-treat participants whether or not randomized treatment (frozen solution) was administered. Intent-to-treat Population comprised of all randomized participants whether or not randomized treatment was administered.
Time Frame: Up to 48 weeks
Population: Efficacy Population. Data is not presented for 'GSK2857916 3.4 mg/kg (Lyophilized)' arm as it is not included in Efficacy Population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid)
Number analyzed (Participants) | 64 | 66
Percentage of Participants | 30 [18.9 to 42.4] | 30 [19.6 to 42.9]

3. Secondary Outcome: Overall Response Rate by Investigator Assessment (IA) (Full Analysis Population)
Description: ORR was determined by the investigator according to the 2016 IMWG response criteria. ORR was calculated as the percentage of participants with a confirmed PR or better (i.e., PR, VGPR, CR and sCR). Confidence intervals were based on the exact method. Percentage values are rounded off.
Time Frame: Up to 186 weeks
Population: Full Analysis Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 97 | 99 | 25
Percentage of Participants | 33 [23.8 to 43.3] | 32 [23.3 to 42.5] | 52 [31.3 to 72.2]

4. Secondary Outcome: Overall Response Rate by Investigator Assessment (Efficacy Population)
Description: as for outcome 3
Time Frame: Up to 186 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid)
Number analyzed (Participants) | 64 | 66
Percentage of Participants | 33 [21.6 to 45.7] | 26 [15.8 to 38.0]

5. Secondary Outcome: Clinical Benefit Rate (CBR) by Investigator Assessment (Full Analysis Population)
Description: CBR was determined by the investigator according to the 2016 IMWG response criteria. CBR was calculated as the percentage of participants with a confirmed minimal response (MR) or better (i.e., MR, PR, VGPR, CR and sCR). Confidence intervals were based on the exact method. Percentage values are rounded off.
Time Frame: Up to 186 weeks
Population: Full Analysis Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 97 | 99 | 25
Percentage of Participants | 35 [25.6 to 45.4] | 38 [28.8 to 48.7] | 60 [38.7 to 78.9]

6. Secondary Outcome: Clinical Benefit Rate by Investigator Assessment (Efficacy Population)
Description: CBR was determined by the investigator according to the 2016 IMWG response criteria. CBR was calculated as the percentage of participants with a confirmed MR or better (i.e., MR, PR, VGPR, CR and sCR). Confidence intervals were based on the exact method. Percentage values are rounded off.
Time Frame: Up to 186 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid)
Number analyzed (Participants) | 64 | 66
Percentage of Participants | 34 [22.9 to 47.3] | 35 [23.5 to 47.6]

7. Secondary Outcome: Clinical Benefit Rate by Independent Review Committee (Full Analysis Population)
Description: CBR was determined according to the 2016 IMWG response criteria by IRC. CBR was calculated as the percentage of participants with a confirmed MR or better (i.e., MR, PR, VGPR, CR and sCR). Confidence intervals were based on the exact method. Percentage values are rounded off.
Time Frame: Up to 186 weeks
Population: Full Analysis Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 97 | 99 | 25
Percentage of Participants | 36 [26.6 to 46.5] | 40 [30.7 to 50.7] | 56 [34.9 to 75.6]

8. Secondary Outcome: Clinical Benefit Rate by Independent Review Committee (Efficacy Population)
Description: as for outcome 7
Time Frame: Up to 186 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid)
Number analyzed (Participants) | 64 | 66
Percentage of Participants | 34 [22.9 to 47.3] | 38 [26.2 to 50.7]

9. Secondary Outcome: Duration of Response (DoR) by Investigator Assessment (Full Analysis Population)
Description: DoR is defined as the time from first documented evidence of PR or better until the earliest date of documented disease progression (PD) per IMWG response criteria; or death due to PD among participants who achieved an overall response, i.e., confirmed PR or better. DOR based on responses assessed by investigator is presented. Median and inter-quartile range (first quartile and third quartile) of DOR are presented.
Time Frame: Up to 186 weeks
Population: Full Analysis Population. Only responders (confirmed PR or better) by investigator assessment were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 32 | 32 | 13
Months | 12.4 [4.2 to 21.4] | 12.6 [5.6 to 22.8] | 5.3 [2.8 to 9.0]

10. Secondary Outcome: Duration of Response by Investigator Assessment (Efficacy Population)
Description: DoR is defined as the time from first documented evidence of PR or better until the earliest date of documented PD per IMWG response criteria; or death due to PD among participants who achieved an overall response, i.e., confirmed PR or better. DOR based on responses assessed by investigator is presented. Median and inter-quartile range (first quartile and third quartile) of DOR are presented.
Time Frame: Up to 186 weeks
Population: Efficacy Population. Data is not presented for 'GSK2857916 3.4 mg/kg (Lyophilized)' arm as it is not included in Efficacy Population. Only responders (confirmed PR or better) by investigator assessment were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid)
Number analyzed (Participants) | 21 | 17
Months | 6.9 [4.2 to 20.8] | 15.9 [12.6 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived

11. Secondary Outcome: Duration of Response by Independent Review Committee (Full Analysis Population)
Description: DoR is defined as the time from first documented evidence of PR or better until the earliest date of documented PD per IMWG response criteria; or death due to PD among participants who achieved an overall response, i.e., confirmed PR or better. DOR based on responses assessed by IRC is presented. Median and inter-quartile range (first quartile and third quartile) of DOR are presented.
Time Frame: Up to 186 weeks
Population: Full Analysis Population. Only responders (confirmed PR or better) by Independent Review Committee were included in this analysis
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 31 | 35 | 13
Months | 12.5 [4.2 to 19.4] | 6.2 [4.2 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. | 9.0 [3.4 to 10.4]

12. Secondary Outcome: Duration of Response by Independent Review Committee (Efficacy Population)
Description: as for outcome 11
Time Frame: Up to 186 weeks
Population: Efficacy Population. Data is not presented for 'GSK2857916 3.4 mg/kg (Lyophilized)' arm as it is not included in Efficacy Population. Only responders (confirmed PR or better) by Independent Review Committee were included in this analysis
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid)
Number analyzed (Participants) | 20 | 20
Months | 11.0 [4.0 to 19.4] | 15.9 [4.2 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.

13. Secondary Outcome: Time to Response by Investigator Assessment (Full Analysis Population)
Description: Time to response is defined as the time between the date of randomization and the first documented evidence of response (PR or better), among participants who achieve a response (i.e., confirmed PR or better). Time to response based on responses assessed by investigator is presented. Median and inter-quartile range (first quartile and third quartile) of time to response are presented.
Time Frame: Up to 186 weeks
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 32 | 32 | 13
Months | 1.5 [0.8 to 2.5] | 1.5 [0.9 to 3.0] | 0.9 [0.8 to 1.0]

14. Secondary Outcome: Time to Response by Investigator Assessment (Efficacy Population)
Description: as for outcome 13
Time Frame: Up to 186 weeks
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid)
Number analyzed (Participants) | 21 | 17
Months | 1.4 [0.8 to 2.8] | 1.5 [1.4 to 2.8]

15. Secondary Outcome: Time to Response by Independent Review Committee (Full Analysis Population)
Description: Time to response is defined as the time between the date of randomization and the first documented evidence of response (PR or better), among participants who achieve a response (i.e., confirmed PR or better). Time to response based on responses assessed by IRC is presented. Median and inter-quartile range (first quartile and third quartile) of time to response are presented.
Time Frame: Up to 186 weeks
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 31 | 35 | 13
Months | 1.5 [0.8 to 2.2] | 1.4 [0.8 to 2.8] | 0.9 [0.8 to 2.3]

16. Secondary Outcome: Time to Response by Independent Review Committee (Efficacy Population)
Description: as for outcome 15
Time Frame: Up to 186 weeks
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid)
Number analyzed (Participants) | 20 | 20
Months | 1.5 [0.8 to 2.5] | 1.4 [1.1 to 1.9]

17. Secondary Outcome: Progression Free Survival by Investigator Assessment
Description: Progression free survival is defined as the time from randomization until the earliest date of documented PD per IMWG, or death due to any cause. Progressive Disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. Progression free survival based on responses assessed by investigator is presented. Median and inter-quartile range (first quartile and third quartile) of progression free survival are presented.
Time Frame: Up to 186 weeks
Population: Full Analysis Population
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 97 | 99 | 25
Months | 2.2 [0.8 to 7.7] | 3.2 [1.0 to 9.8] | 3.6 [1.5 to 8.7]

18. Secondary Outcome: Progression Free Survival by Independent Review Committee
Description: Progression free survival is defined as the time from randomization until the earliest date of documented PD per IMWG, or death due to any cause. Progressive Disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. Progression free survival based on responses assessed by IRC is presented. Median and inter-quartile range (first quartile and third quartile) of progression free survival are presented.
Time Frame: Up to 186 weeks
Population: Full Analysis Population
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 97 | 99 | 25
Months | 2.8 [0.9 to 9.7] | 3.9 [0.8 to 9.0] | 5.7 [2.2 to 9.7]

19. Secondary Outcome: Time to Progression by Investigator Assessment
Description: Time to progression is defined as the time from randomization until the earliest date of documented PD per IMWG, or death due to PD. Time to Progression based on responses assessed by investigator is presented. Median and inter-quartile range (first quartile and third quartile) of time to progression are presented.
Time Frame: Up to 186 weeks
Population: Full Analysis Population
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 97 | 99 | 25
Months | 2.2 [0.8 to 7.7] | 3.9 [1.0 to 11.9] | 3.6 [1.5 to 9.7]

20. Secondary Outcome: Time to Progression by Independent Review Committee
Description: Time to progression is defined as the time from randomization until the earliest date of documented PD per IMWG, or death due to PD. Time to Progression based on responses assessed by IRC is presented. Median and inter-quartile range (first quartile and third quartile) of time to progression are presented.
Time Frame: Up to 186 weeks
Population: Full Analysis Population
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 97 | 99 | 25
Months | 2.9 [0.9 to 9.7] | 4.9 [0.8 to 11.1] | 5.7 [2.2 to 9.7]

21. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization until death due to any cause. Overall survival was analyzed using the Kaplan-Meier method by dose level. Median and inter-quartile range (first quartile and third quartile) of overall survival are presented.
Time Frame: Up to 186 weeks
Population: Full Analysis Population
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 97 | 99 | 25
Months | 15.3 [4.8 to 36.4] | 14.0 [6.2 to 26.6] | 24.5 [7.7 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.

22. Secondary Outcome: Number of Participants With Change From Baseline in Hematology Parameters With Respect to the Normal Range
Description: Following parameters were assessed:basophils,eosinophils,hematocrit,mean corpuscular hemoglobin (MCH),MCH concentration,MC volume,monocyte,erythrocytes, reticulocytes.Baseline is latest pre-dose assessment(Day1)with a non-missing value, including unscheduled visits.Data was categorized as decrease to low(value below lower limit of normal range[LNR]),increase to high(value above upper LNR),change to normal/no change(NC).If values were unchanged(eg.high to high) or whose value became normal,were recorded in change to normal/NC category.Participants were counted twice if participant had both decreased to low/increased to high during post-Baseline(PB).Data for worst case PB is presented.Full Safety Population(FSP) comprised of all participants who received at least 1dose of study drug(frozen liquid or lyophilized powder). 3 out of 221 participants did not receive any study treatment and thus, were excluded from the Full Safety Population.
Time Frame: Baseline (Day 1) and Up to 186 weeks
Population: Full Safety Population. All the participants in the study were included in the analysis (95, 99 and 24 Participants), but only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Participants
  Basophils, decrease to low, n=94,96,23: number analyzed (Participants) | 94 | 96 | 23
  Basophils, decrease to low, n=94,96,23 | 2 | 7 | 0
  Basophils, change to normal or NC, n=94,96,23: number analyzed (Participants) | 94 | 96 | 23
  Basophils, change to normal or NC, n=94,96,23 | 87 | 85 | 19
  Basophils, increase to high, n=94,96,23: number analyzed (Participants) | 94 | 96 | 23
  Basophils, increase to high, n=94,96,23 | 5 | 5 | 4
  Eosinophils, decrease to low, n=95,97,23: number analyzed (Participants) | 95 | 97 | 23
  Eosinophils, decrease to low, n=95,97,23 | 14 | 13 | 0
  Eosinophils, change to normal or NC, n=95,97,23: number analyzed (Participants) | 95 | 97 | 23
  Eosinophils, change to normal or NC, n=95,97,23 | 71 | 78 | 16
  Eosinophils, increase to high, n=95,97,23: number analyzed (Participants) | 95 | 97 | 23
  Eosinophils, increase to high, n=95,97,23 | 10 | 8 | 7
  Hematocrit, decrease to low, n=95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Hematocrit, decrease to low, n=95,97,24 | 10 | 3 | 1
  Hematocrit, change to normal or NC, n=95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Hematocrit, change to normal or NC, n=95,97,24 | 84 | 94 | 23
  Hematocrit, increase to high, n=95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Hematocrit, increase to high, n=95,97,24 | 3 | 0 | 0
  Mean Corpuscular Hemoglobin, decrease to low, n=95,95,21: number analyzed (Participants) | 95 | 95 | 21
  Mean Corpuscular Hemoglobin, decrease to low, n=95,95,21 | 14 | 17 | 5
  Mean Corpuscular Hemoglobin, change to normal or NC, n=95,95,21: number analyzed (Participants) | 95 | 95 | 21
  Mean Corpuscular Hemoglobin, change to normal or NC, n=95,95,21 | 79 | 68 | 14
  Mean Corpuscular Hemoglobin, increase to high, n=95,95,21: number analyzed (Participants) | 95 | 95 | 21
  Mean Corpuscular Hemoglobin, increase to high, n=95,95,21 | 2 | 12 | 2
  MCH Concentration, decrease to low, n=94,96,21: number analyzed (Participants) | 94 | 96 | 21
  MCH Concentration, decrease to low, n=94,96,21 | 20 | 28 | 6
  MCH Concentration, change to normal or NC, n=94,96,21: number analyzed (Participants) | 94 | 96 | 21
  MCH Concentration, change to normal or NC, n=94,96,21 | 70 | 66 | 14
  MCH Concentration, increase to high, n=94,96,21: number analyzed (Participants) | 94 | 96 | 21
  MCH Concentration, increase to high, n=94,96,21 | 5 | 2 | 1
  Mean Corpuscular Volume, decrease to low, n=95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Mean Corpuscular Volume, decrease to low, n=95,97,24 | 12 | 15 | 4
  Mean Corpuscular Volume, change to normal or NC, n=95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Mean Corpuscular Volume, change to normal or NC, n=95,97,24 | 77 | 73 | 18
  Mean Corpuscular Volume, increase to high, n=95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Mean Corpuscular Volume, increase to high, n=95,97,24 | 7 | 10 | 3
  Monocytes, decrease to low, n=95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Monocytes, decrease to low, n=95,97,24 | 6 | 10 | 1
  Monocytes, change to normal or NC, n=95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Monocytes, change to normal or NC, n=95,97,24 | 62 | 50 | 12
  Monocytes, increase to high, n=95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Monocytes, increase to high, n=95,97,24 | 28 | 45 | 12
  Erythrocytes, decrease to low, n=95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Erythrocytes, decrease to low, n=95,97,24 | 4 | 1 | 0
  Erythrocytes, change to normal or NC, n=95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Erythrocytes, change to normal or NC, n=95,97,24 | 91 | 95 | 21
  Erythrocytes, increase to high, n=95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Erythrocytes, increase to high, n=95,97,24 | 2 | 1 | 3
  Reticulocytes, decrease to low, n=73,65,19: number analyzed (Participants) | 73 | 65 | 19
  Reticulocytes, decrease to low, n=73,65,19 | 11 | 15 | 7
  Reticulocytes, change to normal or NC, n=73,65,19: number analyzed (Participants) | 73 | 65 | 19
  Reticulocytes, change to normal or NC, n=73,65,19 | 49 | 33 | 3
  Reticulocytes, increase to high, n=73,65,19: number analyzed (Participants) | 73 | 65 | 19
  Reticulocytes, increase to high, n=73,65,19 | 16 | 21 | 10

23. Secondary Outcome: Number of Participants With Grade Change From Baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of following hematology parameters: hemoglobin (Hb), lymphocyte count (Lymph), neutrophil count (Neutro), platelet count (PC), and leukocyte count (leuko). The laboratory parameters were graded according to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. An increase is defined as an increase in CTCAE grade relative to Baseline grade. Data for worst-case post Baseline is presented. Only those participants with increase to grade 3 and increase to grade 4 have been presented.
Time Frame: Baseline (Day 1) and Up to 186 weeks
Population: Full Safety Population. 3 participants out of 221 participants did not receive any study treatment and thus, were excluded from the Full Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 97 | 24
Participants
  Hb, Hb increased, increase to Grade 3 | 0 | 0 | 0
  Hb, Hb increased, increase to Grade 4 | 0 | 0 | 0
  Hb, Anemia, increase to Grade 3 | 19 | 30 | 5
  Hb, Anemia, increase to Grade 4 | 0 | 0 | 0
  Lymph, Lymph count increased, increase to Grade 3 | 0 | 0 | 0
  Lymph, Lymph count increased, increase to Grade 4 | 0 | 0 | 0
  Lymph, Lymph count decreased, increase to Grade 3 | 16 | 24 | 6
  Lymph, Lymph count decreased, increase to Grade 4 | 5 | 5 | 2
  Neutro, increase to Grade 3 | 4 | 10 | 2
  Neutro, increase to Grade 4 | 6 | 3 | 1
  PC, increase to Grade 3 | 9 | 11 | 1
  PC, increase to Grade 4 | 13 | 25 | 2
  Leuko, Leukocytosis, increase to Grade 3 | 0 | 0 | 0
  Leuko, Leukocytosis, increase to Grade 4 | 0 | 0 | 0
  Leuko, Leuko decreased, increase to Grade 3 | 5 | 9 | 2
  Leuko, Leuko decreased, increase to Grade 4 | 3 | 3 | 0

24. Secondary Outcome: Number of Participants With Change From Baseline in Clinical Chemistry Parameters With Respect to the Normal Range
Description: Blood samples were collected for analysis of clinical chemistry parameters: bicarbonate, direct bilirubin(D.Bil), calcium, chloride, lactate dehydrogenase(LDH), total protein,Urea enzymatic colorimetry.Baseline is latest pre-dose assessment(Day 1) with a non-missing value, including unscheduled visits. Number of participants with worst case clinical chemistry change from Baseline with respect to normal range are presented. Data was categorized as decrease to low (value below the lower LNR), increase to high (value above the upper LNR) and change to normal or NC. If values were unchanged (example: high to high), or whose value became normal, were recorded in the change to normal or NC category. Participants were counted twice if the participant had both decreased to low and increased to high during post Baseline. 3 out of 221participants did not receive any study treatment, were excluded from FSP.
Time Frame: Baseline (Day 1) and Up to 186 weeks
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Participants
  Bicarbonate, decrease to low, n=90,93,24: number analyzed (Participants) | 90 | 93 | 24
  Bicarbonate, decrease to low, n=90,93,24 | 12 | 22 | 4
  Bicarbonate, change to normal or NC, n=90,93,24: number analyzed (Participants) | 90 | 93 | 24
  Bicarbonate, change to normal or NC, n=90,93,24 | 67 | 59 | 16
  Bicarbonate, increase to high, n=90,93,24: number analyzed (Participants) | 90 | 93 | 24
  Bicarbonate, increase to high, n=90,93,24 | 12 | 16 | 4
  Direct Bilirubin, decrease to low, n=70,72,21: number analyzed (Participants) | 70 | 72 | 21
  Direct Bilirubin, decrease to low, n=70,72,21 | 0 | 2 | 0
  Direct Bilirubin, change to normal or NC, n=70,72,21: number analyzed (Participants) | 70 | 72 | 21
  Direct Bilirubin, change to normal or NC, n=70,72,21 | 60 | 60 | 20
  Direct Bilirubin, increase to high, n=70,72,21: number analyzed (Participants) | 70 | 72 | 21
  Direct Bilirubin, increase to high, n=70,72,21 | 10 | 10 | 1
  Calcium, decrease to low, n=95,98,24: number analyzed (Participants) | 95 | 98 | 24
  Calcium, decrease to low, n=95,98,24 | 26 | 28 | 8
  Calcium, change to normal or NC, n=95,98,24: number analyzed (Participants) | 95 | 98 | 24
  Calcium, change to normal or NC, n=95,98,24 | 49 | 48 | 9
  Calcium, increase to high, n=95,98,24: number analyzed (Participants) | 95 | 98 | 24
  Calcium, increase to high, n=95,98,24 | 29 | 27 | 9
  Chloride, decrease to low, n=94,97,24: number analyzed (Participants) | 94 | 97 | 24
  Chloride, decrease to low, n=94,97,24 | 17 | 14 | 2
  Chloride, change to normal or NC, n=94,97,24: number analyzed (Participants) | 94 | 97 | 24
  Chloride, change to normal or NC, n=94,97,24 | 63 | 63 | 20
  Chloride, increase to high, n=94,97,24: number analyzed (Participants) | 94 | 97 | 24
  Chloride, increase to high, n=94,97,24 | 14 | 24 | 2
  LDH, decrease to low, n=92,98,23: number analyzed (Participants) | 92 | 98 | 23
  LDH, decrease to low, n=92,98,23 | 1 | 1 | 0
  LDH, change to normal or NC, n=92,98,23: number analyzed (Participants) | 92 | 98 | 23
  LDH, change to normal or NC, n=92,98,23 | 46 | 51 | 12
  LDH, increase to high, n=92,98,23: number analyzed (Participants) | 92 | 98 | 23
  LDH, increase to high, n=92,98,23 | 45 | 47 | 11
  Protein, decrease to low, n=94,98,24: number analyzed (Participants) | 94 | 98 | 24
  Protein, decrease to low, n=94,98,24 | 32 | 32 | 8
  Protein, change to normal or NC, n=94,98,24: number analyzed (Participants) | 94 | 98 | 24
  Protein, change to normal or NC, n=94,98,24 | 49 | 58 | 14
  Protein, increase to high, n=94,98,24: number analyzed (Participants) | 94 | 98 | 24
  Protein, increase to high, n=94,98,24 | 17 | 11 | 2
  Urea enzymatic colorimetry , decrease to low, n=90,93,24: number analyzed (Participants) | 90 | 93 | 24
  Urea enzymatic colorimetry , decrease to low, n=90,93,24 | 10 | 13 | 0
  Urea enzymatic colorimetry, change to normal or NC, n=90,93,24: number analyzed (Participants) | 90 | 93 | 24
  Urea enzymatic colorimetry, change to normal or NC, n=90,93,24 | 66 | 56 | 16
  Urea enzymatic colorimetry, increase to high, n=90,93,24: number analyzed (Participants) | 90 | 93 | 24
  Urea enzymatic colorimetry, increase to high, n=90,93,24 | 15 | 26 | 8

25. Secondary Outcome: Number of Participants With Grade Change From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for analysis of:glucose(Gl), albumin, alkaline phosphatase (ALP), alanine aminotransferase(ALT), aspartate aminotransferase(AST), total bilirubin(T.Bil),creatinine kinase (CK),creatinine, gamma glutamyl transferase (GGT),potassium (Pot), magnesium (Mg),sodium (Sod), phosphate (Ph) urate & estimated glomerular filtration rate (eGFR). Values (Hyper and hypo) for Gl, Pot, Mg and Sod is presented. Grading was according to NCI-CTCAE version 4.03. Grade1: mild; Grade2: moderate; Grade3: severe or medically significant; Grade4: life-threatening consequences.Baseline is latest pre-dose assessment(Day 1) with a non-missing value, including unscheduled visits. An increase is defined as an increase in CTCAE grade relative to Baseline grade. Data for worst-case PB is presented.Only those participants with increase to grade3 and increase to grade4 have been presented. 3 out of 221participants did not receive any study treatment, were excluded from FSP.
Time Frame: Baseline (Day 1) and Up to 186 weeks
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Participants
  Gl, Hyper, increase to Grade 3, n=94,95,24: number analyzed (Participants) | 94 | 95 | 24
  Gl, Hyper, increase to Grade 3, n=94,95,24 | 3 | 5 | 0
  Gl, Hyper, increase to Grade 4, n=94,95,24: number analyzed (Participants) | 94 | 95 | 24
  Gl, Hyper, increase to Grade 4, n=94,95,24 | 0 | 0 | 0
  Gl, Hypo, increase to Grade 3, n=94,95,24: number analyzed (Participants) | 94 | 95 | 24
  Gl, Hypo, increase to Grade 3, n=94,95,24 | 0 | 0 | 0
  Gl, Hypo, increase to Grade 4, n=94,95,24: number analyzed (Participants) | 94 | 95 | 24
  Gl, Hypo, increase to Grade 4, n=94,95,24 | 0 | 0 | 0
  Albumin, increase to Grade 3, n=94,98,24: number analyzed (Participants) | 94 | 98 | 24
  Albumin, increase to Grade 3, n=94,98,24 | 4 | 7 | 1
  Albumin, increase to Grade 4, n=94,98,24: number analyzed (Participants) | 94 | 98 | 24
  Albumin, increase to Grade 4, n=94,98,24 | 0 | 0 | 0
  ALP, increase to Grade 3, n=93,97,24: number analyzed (Participants) | 93 | 97 | 24
  ALP, increase to Grade 3, n=93,97,24 | 1 | 0 | 0
  ALP, increase to Grade 4, n=93,97,24: number analyzed (Participants) | 93 | 97 | 24
  ALP, increase to Grade 4, n=93,97,24 | 0 | 0 | 0
  ALT, increase to Grade 3, n=93,97,24: number analyzed (Participants) | 93 | 97 | 24
  ALT, increase to Grade 3, n=93,97,24 | 0 | 0 | 0
  ALT, increase to Grade 4, n=93,97,24: number analyzed (Participants) | 93 | 97 | 24
  ALT, increase to Grade 4, n=93,97,24 | 0 | 0 | 0
  AST, increase to Grade 3, n=93,96,24: number analyzed (Participants) | 93 | 96 | 24
  AST, increase to Grade 3, n=93,96,24 | 3 | 7 | 0
  AST, increase to Grade 4, n=93,96,24: number analyzed (Participants) | 93 | 96 | 24
  AST, increase to Grade 4, n=93,96,24 | 0 | 0 | 0
  T.Bil, increase to Grade 3, n=92,97,23: number analyzed (Participants) | 92 | 97 | 23
  T.Bil, increase to Grade 3, n=92,97,23 | 0 | 0 | 0
  T.Bil, increase to Grade 4, n=92,97,23: number analyzed (Participants) | 92 | 97 | 23
  T.Bil, increase to Grade 4, n=92,97,23 | 0 | 0 | 0
  CK, increase to Grade 3, n= 87,91,24: number analyzed (Participants) | 87 | 91 | 24
  CK, increase to Grade 3, n= 87,91,24 | 1 | 0 | 1
  CK, increase to Grade 4, n= 87,91,24: number analyzed (Participants) | 87 | 91 | 24
  CK, increase to Grade 4, n= 87,91,24 | 2 | 0 | 0
  Creatinine, increase to Grade 3, n= 95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Creatinine, increase to Grade 3, n= 95,97,24 | 4 | 3 | 0
  Creatinine, increase to Grade 4, n= 95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Creatinine, increase to Grade 4, n= 95,97,24 | 1 | 0 | 0
  GGT, increase to Grade 3, n= 91,95,24: number analyzed (Participants) | 91 | 95 | 24
  GGT, increase to Grade 3, n= 91,95,24 | 5 | 11 | 1
  GGT, increase to Grade 4, n= 91,95,24: number analyzed (Participants) | 91 | 95 | 24
  GGT, increase to Grade 4, n= 91,95,24 | 1 | 1 | 0
  Pot, Hyper,increase to Grade 3, n= 95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Pot, Hyper,increase to Grade 3, n= 95,97,24 | 0 | 1 | 0
  Pot, Hyper,increase to Grade 4, n= 95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Pot, Hyper,increase to Grade 4, n= 95,97,24 | 0 | 0 | 0
  Pot, Hypo, increase to Grade 3, n= 95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Pot, Hypo, increase to Grade 3, n= 95,97,24 | 0 | 4 | 1
  Pot, Hypo, increase to Grade 4, n= 95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Pot, Hypo, increase to Grade 4, n= 95,97,24 | 2 | 0 | 0
  Mg, Hyper, increase to Grade 3, n= 91,96,24: number analyzed (Participants) | 91 | 96 | 24
  Mg, Hyper, increase to Grade 3, n= 91,96,24 | 3 | 1 | 0
  Mg, Hyper, increase to Grade 4, n= 91,96,24: number analyzed (Participants) | 91 | 96 | 24
  Mg, Hyper, increase to Grade 4, n= 91,96,24 | 0 | 0 | 0
  Mg, Hypo, increase to Grade 3, n= 91,96,24: number analyzed (Participants) | 91 | 96 | 24
  Mg, Hypo, increase to Grade 3, n= 91,96,24 | 0 | 0 | 0
  Mg, Hypo, increase to Grade 4, n= 91,96,24: number analyzed (Participants) | 91 | 96 | 24
  Mg, Hypo, increase to Grade 4, n= 91,96,24 | 0 | 0 | 0
  Phosphate, increase to Grade 3, n= 90,93,24: number analyzed (Participants) | 90 | 93 | 24
  Phosphate, increase to Grade 3, n= 90,93,24 | 4 | 8 | 2
  Phosphate, increase to Grade 4, n= 90,93,24: number analyzed (Participants) | 90 | 93 | 24
  Phosphate, increase to Grade 4, n= 90,93,24 | 0 | 0 | 0
  Sod, Hyper, increase to Grade 3, n= 95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Sod, Hyper, increase to Grade 3, n= 95,97,24 | 0 | 0 | 0
  Sod, Hyper, increase to Grade 4, n= 95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Sod, Hyper, increase to Grade 4, n= 95,97,24 | 0 | 0 | 0
  Sod, Hypo, increase to Grade 3, n= 95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Sod, Hypo, increase to Grade 3, n= 95,97,24 | 2 | 6 | 1
  Sod, Hypo, increase to Grade 4, n= 95,97,24: number analyzed (Participants) | 95 | 97 | 24
  Sod, Hypo, increase to Grade 4, n= 95,97,24 | 0 | 0 | 0
  Urate, increase to Grade 3, n= 93,96,24: number analyzed (Participants) | 93 | 96 | 24
  Urate, increase to Grade 3, n= 93,96,24 | 0 | 0 | 0
  Urate, increase to Grade 4, n= 93,96,24: number analyzed (Participants) | 93 | 96 | 24
  Urate, increase to Grade 4, n= 93,96,24 | 3 | 5 | 1
  eGFR, increase to Grade 3, n= 84,85,23: number analyzed (Participants) | 84 | 85 | 23
  eGFR, increase to Grade 3, n= 84,85,23 | 8 | 11 | 0
  eGFR, increase to Grade 4, n= 84,85,23: number analyzed (Participants) | 84 | 85 | 23
  eGFR, increase to Grade 4, n= 84,85,23 | 3 | 1 | 0

26. Secondary Outcome: Number of Participants With Abnormal Findings During Physical Examination
Description: Physical examination included assessment of the head, eyes, ears, nose, throat, skin, thyroid, lungs, cardiovascular, abdomen (liver and spleen), lymph nodes, and extremities. This analysis was planned, but data was not collected and captured in the database.
Time Frame: Up to 186 weeks
Population: Full Safety Population. This analysis was planned, but data was not collected and captured in the database.
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Change From Baseline in Pulse Rate
Description: Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Number of participants with worst case change from Baseline in pulse rate is presented. Data is categorized as: pulse rate 'decrease to <60 beats per minute [bpm]', 'increase to >100 bpm' and 'change to normal or no change'. If values were unchanged (example: increase to >100 bpm to increase to >100 bpm), or whose value became normal, were recorded in the 'change to normal or no change' category. Participants were counted twice if the participant had both 'decreased to <60 bpm' and 'increased to >100 bpm' during post Baseline. Data for worst-case post Baseline is presented.
Time Frame: Baseline (Day 1) and Up to 186 weeks
Population: Full Safety Population. 3 participants out of 221 participants did not receive any study treatment and thus, were excluded from the Full Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Participants
  Decrease to <60 | 14 | 17 | 6
  Change to normal or no change | 57 | 55 | 15
  Increase to >100 | 25 | 28 | 3

28. Secondary Outcome: Number of Participants With Change From Baseline in Body Temperature
Description: Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Number of participants with worst case change from Baseline in body temperature are presented. Data is categorized as: body temperature 'decrease to <=35 degrees celsius', 'increase to >=38 degrees celsius' and 'change to normal or no change'. If values were unchanged (example: increase to >=38 to increase to >=38 degrees celsius), or whose value became normal, were recorded in the 'change to normal or no change' category. Participants were counted twice if the participant had both 'decreased to <=35' and 'increased to >=38 degrees celsius' during post Baseline. Data for worst-case post Baseline is presented.
Time Frame: Baseline (Day 1) and Up to 186 weeks
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 98 | 24
Participants
  Decrease to <=35 | 1 | 3 | 0
  Change to normal or no change | 86 | 85 | 21
  Increase to >=38 | 8 | 10 | 3

29. Secondary Outcome: Number of Participants With Grade Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were graded using NCI CTCAE version 4.03. For SBP: Grade 0: <120 millimeter mercury (mmHg); Grade 1: 120-139 mmHg; Grade 2: 140-159 mmHg; Grade 3: >=160 mmHg. For DBP: Grade 0: <80 mmHg; Grade 1: 80-89 mmHg; Grade 2: 90-99 mmHg; Grade 3: >=100 mmHg. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. An increase is defined as an increase in CTCAE grade relative to Baseline grade. Data for worst-case post Baseline is presented. Only those participants with increase to grade 2 and increase to grade 3 have been presented.
Time Frame: Baseline (Day 1) and Up to 186 weeks
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Participants
  SBP, increase to Grade 2 | 29 | 41 | 4
  SBP, increase to Grade 3 | 14 | 22 | 8
  DBP, increase to Grade 2 | 18 | 16 | 2
  DBP, increase to Grade 3 | 9 | 8 | 1

30. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Common (>=5%) Non-serious Adverse Events and Adverse Events of Special Interest (AESI)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function. Adverse events which were not Serious were considered as non-serious adverse events. Number of participants who had SAEs and common (>=5%) non-SAEs are presented. Number of participants with AESI (keratopathy, dry eye events, blurred vision, thrombocytopenia, infusion-related reactions, corneal events and neutropenia) are also presented.
Time Frame: Up to 186 weeks
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Participants
  Common non-SAE | 93 | 96 | 24
  SAE | 43 | 53 | 15
  Keratopathy | 67 | 74 | 23
  Dry eye events | 17 | 25 | 6
  Blurred vision | 24 | 36 | 10
  Thrombocytopenia | 36 | 56 | 10
  Infusion-related reactions | 20 | 16 | 4
  Corneal events | 68 | 76 | 23
  Neutropenia | 14 | 28 | 2

31. Secondary Outcome: Number of Participants With Change From Baseline in Best Corrected Visual Acuity (BCVA) Test Scores
Description: Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. BCVA score was assessed individually for each eye. BCVA test scores were categorized as no change/improved vision, possible worsened vision and definite worsened vision. No change/improved vision was defined as a change from Baseline <0.12 Logarithm of the Minimum Angle of Resolution (logMAR) score; a possible worsened vision was defined as a change from Baseline >=0.12 to <0.3 logMAR score; a definite worsened vision was defined as a change from Baseline >=0.3 logMAR score. Data for worst-case change from Baseline is presented. 3 participants out of 221 participants did not receive any study treatment and thus, were excluded from the Full Safety Population.
Time Frame: Baseline (Day 1) and Up to 186 weeks
Population: Full Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 88 | 94 | 24
Participants
  Left eye, no change/improved vision, n=88,94,24 | 35 | 45 | 4
  Left eye, possible worsened vision, n=88,94,24 | 11 | 15 | 4
  Left eye, definite worsened vision, n=88,94,24 | 42 | 34 | 16
  Right eye, no change/improved vision, n=87,93,23: number analyzed (Participants) | 87 | 93 | 23
  Right eye, no change/improved vision, n=87,93,23 | 32 | 38 | 5
  Right eye, possible worsened vision, n=87,93,23: number analyzed (Participants) | 87 | 93 | 23
  Right eye, possible worsened vision, n=87,93,23 | 21 | 13 | 6
  Right eye, definite worsened vision, n=87,93,23: number analyzed (Participants) | 87 | 93 | 23
  Right eye, definite worsened vision, n=87,93,23 | 34 | 42 | 12

32. Secondary Outcome: Number of Participants With Intraocular Pressure (IOP) >=22 mmHg Anytime Post-Baseline
Description: Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. IOP was assessed individually for each eye. Number of participants with IOP >=22 mmHg anytime post-Baseline are presented. 3 participants out of 221 participants did not receive any study treatment and thus, were excluded from the Full Safety Population.
Time Frame: Up to 186 weeks
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 88 | 93 | 24
Participants
  Right eye, n=88,93,23: number analyzed (Participants) | 88 | 93 | 23
  Right eye, n=88,93,23 | 17 | 16 | 8
  Left eye, n=88,92,24: number analyzed (Participants) | 88 | 92 | 24
  Left eye, n=88,92,24 | 14 | 15 | 7

33. Secondary Outcome: Number of Participants With Shift in Pupillary Examination Findings From Normal (Baseline) to Abnormal (Worst Post-Baseline)
Description: Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Number of participants with shift in pupillary examination findings from normal (Baseline) to abnormal (worst post-Baseline) are presented.
Time Frame: Baseline and Up to 186 weeks
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 91 | 90 | 23
Participants | 4 | 12 | 3

34. Secondary Outcome: Number of Participants With Shift in Extraocular Muscle Movement From Yes (Baseline) to no (Worst Post-Baseline)
Description: Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Extraocular muscle movement was assessed individually for each eye. Number of participants with shift in extraocular muscle movement from yes (Baseline) to no (worst post-Baseline) are presented. 3 participants out of 221 participants did not receive any study treatment and thus, were excluded from the Full Safety Population.
Time Frame: Baseline and Up to 186 weeks
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 93 | 23
Participants
  Right eye,n=95,93,23 | 0 | 4 | 0
  Left eye,n=93,92,22: number analyzed (Participants) | 93 | 92 | 22
  Left eye,n=93,92,22 | 0 | 2 | 0

35. Secondary Outcome: Number of Participants With Shift in Corneal Epithelium Findings From Normal (Baseline) to Abnormal (Worst Post-Baseline) for Corneal Epithelium (CE) and Corneal Stroma (CS)
Description: Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Corneal epithelium findings for CE and CS were assessed individually for each eye. Number of participants with shift in corneal epithelium findings from normal (Baseline) to abnormal (worst post-Baseline) for CE and CS are presented. 3 participants out of 221 participants did not receive any study treatment and thus, were excluded from the Full Safety Population.
Time Frame: Baseline and Up to 186 weeks
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 92 | 94 | 24
Participants
  CE, Right eye, n=53,54,17: number analyzed (Participants) | 53 | 54 | 17
  CE, Right eye, n=53,54,17 | 39 | 40 | 16
  CE, Left eye,n=55,55,15: number analyzed (Participants) | 55 | 55 | 15
  CE, Left eye,n=55,55,15 | 39 | 44 | 14
  CS, Right eye,n=92,94,24 | 5 | 7 | 3
  CS, Left eye,n=92,89,23: number analyzed (Participants) | 92 | 89 | 23
  CS, Left eye,n=92,89,23 | 8 | 5 | 3

36. Secondary Outcome: Number of Participants With Shift in Corneal Epithelium Findings From no (Baseline) to Yes (Worst Post-Baseline)
Description: Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Corneal epithelium findings like active edema, active opacity, corneal neovascularization (CN), corneal ulcer, epithelial microcystic edema (EME) and subepithelial were performed using a slit lamp. Number of participants with shift in corneal epithelium findings from no (Baseline) to yes (worst post-Baseline) are presented. 3 participants out of 221 participants did not receive any study treatment and thus, were excluded from the Full Safety Population.
Time Frame: Baseline and Up to 186 weeks
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Participants
  Active edema, Right eye, n=94,99,24: number analyzed (Participants) | 94 | 99 | 24
  Active edema, Right eye, n=94,99,24 | 3 | 5 | 1
  Active edema, Left eye,n=95,99,24 | 4 | 4 | 1
  Active opacity, Right eye,n=93,97,24: number analyzed (Participants) | 93 | 97 | 24
  Active opacity, Right eye,n=93,97,24 | 3 | 3 | 3
  Active opacity, Left eye,n=94,95,24: number analyzed (Participants) | 94 | 95 | 24
  Active opacity, Left eye,n=94,95,24 | 4 | 4 | 3
  Corneal Neovascularization, Right eye,n=93,99,24: number analyzed (Participants) | 93 | 99 | 24
  Corneal Neovascularization, Right eye,n=93,99,24 | 1 | 1 | 1
  Corneal Neovascularization, Left eye,n=93,99,23: number analyzed (Participants) | 93 | 99 | 23
  Corneal Neovascularization, Left eye,n=93,99,23 | 1 | 0 | 1
  Corneal ulcer, Right eye,n=61,60,22: number analyzed (Participants) | 61 | 60 | 22
  Corneal ulcer, Right eye,n=61,60,22 | 1 | 1 | 0
  Corneal ulcer, Left eye,n=63,61,20: number analyzed (Participants) | 63 | 61 | 20
  Corneal ulcer, Left eye,n=63,61,20 | 1 | 2 | 0
  Epithelial Microcystic Edema, Right eye,n=95,99,24 | 15 | 24 | 9
  Epithelial Microcystic Edema, Left eye,n=95,99,23: number analyzed (Participants) | 95 | 99 | 23
  Epithelial Microcystic Edema, Left eye,n=95,99,23 | 16 | 25 | 8
  Subepithelial haze, Right eye,n=95,98,24: number analyzed (Participants) | 95 | 98 | 24
  Subepithelial haze, Right eye,n=95,98,24 | 18 | 28 | 8
  Subepithelial haze, Left eye,n=95,97,23: number analyzed (Participants) | 95 | 97 | 23
  Subepithelial haze, Left eye,n=95,97,23 | 18 | 29 | 6

37. Secondary Outcome: Number of Participants With Shift in Tear Break-up Time From >10 Seconds (Baseline) to <=5 Seconds (Worst Post-Baseline)
Description: Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Number of participants with shift in tear break-up time from >10 seconds (Baseline) to <=5 seconds (worst post-Baseline) are presented. 3 participants out of 221 participants did not receive any study treatment and thus, were excluded from the Full Safety Population.
Time Frame: Baseline and Up to 186 weeks
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 34 | 31 | 2
Participants
  Left eye,n=34,30,2: number analyzed (Participants) | 34 | 30 | 2
  Left eye,n=34,30,2 | 14 | 12 | 2
  Right eye,n=30,31,2: number analyzed (Participants) | 30 | 31 | 2
  Right eye,n=30,31,2 | 11 | 12 | 1

38. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC[0-infinity]) of GSK2857916 Following IV Dose in Participants With RRMM
Description: Blood samples were collected at designated timepoints. Pharmacokinetic (PK) parameters of GSK2857916 were calculated using non-compartmental methods. Full Pharmacokinetic (PK) Population comprised of all participants in the Full Safety Population who had atleast 1 non-missing PK assessment.
Time Frame: Cycle 1 and Cycle 3: Pre-dose, end of infusion (EOI), 2 hours and 24 hours post start of infusion (SOI) on Day 1, anytime on Day 4, and anytime on Day 8 to Day 15 (each cycle of 21 days)
Population: Full PK Population. All the participants in the study were included in the analysis (95, 99 and 24 Participants), but only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours*microgram per milliliter
  Cycle 1,n=26,18,18: number analyzed (Participants) | 26 | 18 | 18
  Cycle 1,n=26,18,18 | 5644 (39.6) | 6495 (54.3) | 6962 (51.4)
  Cycle 3, n=19,21,9: number analyzed (Participants) | 19 | 21 | 9
  Cycle 3, n=19,21,9 | 7848 (42.7) | 9199 (45.1) | 9694 (49.9)

39. Secondary Outcome: Area Under the Concentration-time Curve Over the Dosing Interval (AUC[0-tau]) of GSK2857916 Following IV Dose in Participants With RRMM
Description: Blood samples were collected at designated timepoints. PK parameters of GSK2857916 were calculated using non-compartmental methods.
Time Frame: Cycle 1 and Cycle 3: Pre-dose, EOI, 2 hours and 24 hours post SOI on Day 1, anytime on Day 4, and anytime on Day 8 to Day 15 (each cycle of 21 days)
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours*microgram per milliliter
  Cycle 1, n=30,20,22: number analyzed (Participants) | 30 | 20 | 22
  Cycle 1, n=30,20,22 | 4666 (45.7) | 5678 (40.1) | 5946 (37.2)
  Cycle 3, n=26,24,11: number analyzed (Participants) | 26 | 24 | 11
  Cycle 3, n=26,24,11 | 6399 (31.6) | 6941 (34.2) | 7593 (34.5)

40. Secondary Outcome: Area Under the Concentration-time Curve From Zero to Time of Last Quantifiable Concentration (AUC[0-tlast]) of GSK2857916 Following IV Dose in Participants With RRMM
Description: as for outcome 39
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours*microgram per milliliter
  Cycle 1, n=32,21,22: number analyzed (Participants) | 32 | 21 | 22
  Cycle 1, n=32,21,22 | 4607 (54.4) | 5567 (51.0) | 6293 (45.7)
  Cycle 3, n=28,28,11: number analyzed (Participants) | 28 | 28 | 11
  Cycle 3, n=28,28,11 | 6033 (44.7) | 6084 (73.8) | 8388 (46.1)

41. Secondary Outcome: Maximum Observed Concentration (Cmax) of GSK2857916 Following IV Dose in Participants With RRMM
Description: as for outcome 39
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Microgram per milliliter
  Cycle 1, n=32,21,22: number analyzed (Participants) | 32 | 21 | 22
  Cycle 1, n=32,21,22 | 42.51 (26.3) | 52.03 (19.8) | 51.32 (18.3)
  Cycle 3, n=29,28,11: number analyzed (Participants) | 29 | 28 | 11
  Cycle 3, n=29,28,11 | 42.35 (25.6) | 45.5 (25.3) | 48.06 (17.1)

42. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of GSK2857916 Following IV Dose in Participants With RRMM
Description: as for outcome 39
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours
  Cycle 1, n=32,21,22: number analyzed (Participants) | 32 | 21 | 22
  Cycle 1, n=32,21,22 | 0.780 [0.42 to 2.50] | 0.700 [0.43 to 2.15] | 0.750 [0.48 to 2.88]
  Cycle 3, n=29,28,11: number analyzed (Participants) | 29 | 28 | 11
  Cycle 3, n=29,28,11 | 0.580 [0.47 to 2.03] | 0.715 [0.42 to 2.90] | 0.870 [0.50 to 2.02]

43. Secondary Outcome: Terminal Half-life (t1/2) of GSK2857916 Following IV Dose in Participants With RRMM
Description: as for outcome 39
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours
  Cycle 1, n=29,19,22: number analyzed (Participants) | 29 | 19 | 22
  Cycle 1, n=29,19,22 | 164.4 (46.2) | 165.8 (55.0) | 196.2 (40.9)
  Cycle 3, n=26,23,11: number analyzed (Participants) | 26 | 23 | 11
  Cycle 3, n=26,23,11 | 193.7 (48.4) | 214.4 (45.9) | 279.5 (40.3)

44. Secondary Outcome: AUC(0-infinity) of GSK2857916 Total Antibody Following IV Dose in Participants With RRMM
Description: Blood samples were collected at designated timepoints. PK parameters of GSK2857916 total antibody were calculated using non-compartmental methods.
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours*microgram per milliliter
  Cycle 1, n=16,10,9: number analyzed (Participants) | 16 | 10 | 9
  Cycle 1, n=16,10,9 | 10268 (65.8) | 10209 (64.9) | 10170 (75.0)
  Cycle 3, n=10,11,3: number analyzed (Participants) | 10 | 11 | 3
  Cycle 3, n=10,11,3 | 20526 (45.1) | 18637 (69.4) | 22782 (161.1)

45. Secondary Outcome: AUC(0-tau) of GSK2857916 Total Antibody Following IV Dose in Participants With RRMM
Description: as for outcome 44
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours*microgram per milliliter
  Cycle 1, n=29,18,19: number analyzed (Participants) | 29 | 18 | 19
  Cycle 1, n=29,18,19 | 7305 (41.9) | 9566 (42.2) | 9029 (40.2)
  Cycle 3, n=23,24,11: number analyzed (Participants) | 23 | 24 | 11
  Cycle 3, n=23,24,11 | 11243 (34.6) | 11646 (38.0) | 15311 (43.9)

46. Secondary Outcome: AUC(0-tlast) of GSK2857916 Total Antibody Following IV Dose in Participants With RRMM
Description: as for outcome 44
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours*microgram per milliliter
  Cycle 1, n=30,19,20: number analyzed (Participants) | 30 | 19 | 20
  Cycle 1, n=30,19,20 | 7417 (58.5) | 9628 (52.8) | 9017 (55.4)
  Cycle 3, n=27,26,11: number analyzed (Participants) | 27 | 26 | 11
  Cycle 3, n=27,26,11 | 10725 (59.4) | 11295 (80.0) | 17715 (61.0)

47. Secondary Outcome: Cmax of GSK2857916 Total Antibody Following IV Dose in Participants With RRMM
Description: as for outcome 44
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Microgram per milliliter
  Cycle 1, n=30,19,20: number analyzed (Participants) | 30 | 19 | 20
  Cycle 1, n=30,19,20 | 48.94 (30.0) | 61.06 (26.9) | 60.08 (18.3)
  Cycle 3, n=29,28,11: number analyzed (Participants) | 29 | 28 | 11
  Cycle 3, n=29,28,11 | 49.34 (32.9) | 55.60 (26.5) | 65.07 (17.4)

48. Secondary Outcome: Tmax of GSK2857916 Total Antibody Following IV Dose in Participants With RRMM
Description: as for outcome 44
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours
  Cycle 1, n=30,19,20: number analyzed (Participants) | 30 | 19 | 20
  Cycle 1, n=30,19,20 | 1.750 [0.42 to 2.50] | 1.870 [0.50 to 24.50] | 0.650 [0.48 to 2.17]
  Cycle 3, n=29,28,11: number analyzed (Participants) | 29 | 28 | 11
  Cycle 3, n=29,28,11 | 0.830 [0.47 to 46.05] | 1.150 [0.42 to 2.90] | 1.750 [0.50 to 2.02]

49. Secondary Outcome: t1/2 of GSK2857916 Total Antibody Following IV Dose in Participants With RRMM
Description: as for outcome 44
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours
  Cycle 1, n=29,17,19: number analyzed (Participants) | 29 | 17 | 19
  Cycle 1, n=29,17,19 | 241.8 (49.3) | 250.8 (70.3) | 299.8 (61.0)
  Cycle 3, n=23,23,11: number analyzed (Participants) | 23 | 23 | 11
  Cycle 3, n=23,23,11 | 352.4 (52.6) | 372.0 (49.6) | 557.3 (91.7)

50. Secondary Outcome: AUC(0-infinity) of Cysteine-maleimidocaproyl Monomethyl Auristatin F (Cys-mcMMAF) Following IV Dose of GSK2857916 in Participants With RRMM
Description: Blood samples were collected at designated timepoints. PK parameters of Cys-mcMMAF were calculated using non-compartmental methods.
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours*nanogram per milliliter
  Cycle 1, n=27,20,19: number analyzed (Participants) | 27 | 20 | 19
  Cycle 1, n=27,20,19 | NA (NA) — Cys-mcMMAF was not detectable throughout the elimination phase; therefore, AUC(0-infinity) could not be estimated. | NA (NA) — Cys-mcMMAF was not detectable throughout the elimination phase; therefore, AUC(0-infinity) could not be estimated. | NA (NA) — Cys-mcMMAF was not detectable throughout the elimination phase; therefore, AUC(0-infinity) could not be estimated.
  Cycle 3, n=26,29,11: number analyzed (Participants) | 26 | 29 | 11
  Cycle 3, n=26,29,11 | NA (NA) — Cys-mcMMAF was not detectable throughout the elimination phase; therefore, AUC(0-infinity) could not be estimated. | NA (NA) — Cys-mcMMAF was not detectable throughout the elimination phase; therefore, AUC(0-infinity) could not be estimated. | NA (NA) — Cys-mcMMAF was not detectable throughout the elimination phase; therefore, AUC(0-infinity) could not be estimated.

51. Secondary Outcome: AUC(0-tau) of Cys-mcMMAF Following IV Dose of GSK2857916 in Participants With RRMM
Description: as for outcome 50
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours*nanogram per milliliter
  Cycle 1, n=27,20,19: number analyzed (Participants) | 27 | 20 | 19
  Cycle 1, n=27,20,19 | NA (NA) — Cys-mcMMAF was not detectable throughout the dosing interval; therefore, AUC(0-tau) could not be estimated. | NA (NA) — Cys-mcMMAF was not detectable throughout the dosing interval; therefore, AUC(0-tau) could not be estimated. | NA (NA) — Cys-mcMMAF was not detectable throughout the dosing interval; therefore, AUC(0-tau) could not be estimated.
  Cycle 3, n=26,29,11: number analyzed (Participants) | 26 | 29 | 11
  Cycle 3, n=26,29,11 | NA (NA) — Cys-mcMMAF was not detectable throughout the dosing interval; therefore, AUC(0-tau) could not be estimated. | NA (NA) — Cys-mcMMAF was not detectable throughout the dosing interval; therefore, AUC(0-tau) could not be estimated. | NA (NA) — Cys-mcMMAF was not detectable throughout the dosing interval; therefore, AUC(0-tau) could not be estimated.

52. Secondary Outcome: AUC(0-tlast) of Cysteine-maleimidocaproyl Monomethyl Auristatin F (Cys-mcMMAF) Following IV Dose of GSK2857916 in Participants With RRMM
Description: as for outcome 50
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours*nanogram per milliliter
  Cycle 1, n=27,20,19: number analyzed (Participants) | 27 | 20 | 19
  Cycle 1, n=27,20,19 | 79.26 (61.0) | 113.57 (58.3) | 100.35 (51.8)
  Cycle 3, n=26,29,11: number analyzed (Participants) | 26 | 29 | 11
  Cycle 3, n=26,29,11 | 70.84 (46.9) | 74.04 (73.0) | 69.83 (36.6)

53. Secondary Outcome: Cmax of Cys-mcMMAF Following IV Dose of GSK2857916 in Participants With RRMM
Description: as for outcome 50
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Nanogram per milliliter
  Cycle 1, n=27,20,19: number analyzed (Participants) | 27 | 20 | 19
  Cycle 1, n=27,20,19 | 0.903 (63.9) | 1.148 (64.7) | 1.017 (61.4)
  Cycle 3, n=26,29,11: number analyzed (Participants) | 26 | 29 | 11
  Cycle 3, n=26,29,11 | 0.660 (52.3) | 0.749 (66.2) | 0.656 (47.6)

54. Secondary Outcome: Tmax of Cys-mcMMAF Following IV Dose of GSK2857916 in Participants With RRMM
Description: as for outcome 50
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours
  Cycle 1, n=27,20,19: number analyzed (Participants) | 27 | 20 | 19
  Cycle 1, n=27,20,19 | 22.830 [1.92 to 65.63] | 23.835 [17.38 to 72.65] | 24.080 [0.97 to 69.47]
  Cycle 3, n=26,29,11: number analyzed (Participants) | 26 | 29 | 11
  Cycle 3, n=26,29,11 | 23.235 [0.58 to 46.08] | 22.570 [0.55 to 70.98] | 22.780 [0.50 to 71.93]

55. Secondary Outcome: t1/2 of Cys-mcMMAF Following IV Dose of GSK2857916 in Participants With RRMM
Description: as for outcome 50
Time Frame: as for outcome 39
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 95 | 99 | 24
Hours
  Cycle 1, n=27,20,19: number analyzed (Participants) | 27 | 20 | 19
  Cycle 1, n=27,20,19 | NA (NA) — Cys-mcMMAF was not detectable throughout the elimination phase; therefore, t1/2 could not be estimated. | NA (NA) — Cys-mcMMAF was not detectable throughout the elimination phase; therefore, t1/2 could not be estimated. | NA (NA) — Cys-mcMMAF was not detectable throughout the elimination phase; therefore, t1/2 could not be estimated.
  Cycle 3, n=26,29,11: number analyzed (Participants) | 26 | 29 | 11
  Cycle 3, n=26,29,11 | NA (NA) — Cys-mcMMAF was not detectable throughout the elimination phase; therefore, t1/2 could not be estimated. | NA (NA) — Cys-mcMMAF was not detectable throughout the elimination phase; therefore, t1/2 could not be estimated. | NA (NA) — Cys-mcMMAF was not detectable throughout the elimination phase; therefore, t1/2 could not be estimated.

56. Secondary Outcome: Number of Participants With at Least One Confirmed Positive Post-Baseline Anti-drug Antibody (ADA) Result
Description: Serum samples were collected for the determination of anti-GSK2857916 antibodies (ADA) using a validated electrochemiluminescent (ECL) immunoassay. The assay involved screening, confirmation and titration steps. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for the specificity using the confirmation assay. Samples that confirmed positive in the confirmation assay were reported as 'positive'. Confirmed positive ADA samples were further characterized in the titration assay to quasi-quantitate the amount of ADA in the sample. Additionally, confirmed positive ADA samples were also tested in a validated neutralizing antibody assay to determine the potential neutralizing activity of the ADA.
Time Frame: Up to 186 weeks
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 89 | 92 | 24
Participants | 2 | 0 | 0

57. Secondary Outcome: Titers of Anti-drug Antibodies Against GSK2857916
Description: Serum samples were collected for the determination of ADA using a validated ECL immunoassay. The assay involved screening, confirmation and titration steps. If serum samples contained ADA, they were further analyzed for the specificity of antibodies by a confirmation assay. Confirmed positive samples were titrated to obtain the titers of antibodies. Titers of anti-drug antibodies against GSK2857916 is presented. No participant was found with positive results for ADA test in arm GSK2857916 3.4 mg/kg (Lyophilized). Hence, titer values was not presented for the arm.
Time Frame: Up to 186 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Titers
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 4 | 2 | 0
Titers | 125.0 (50.00) | 100.0 (0.00) |

58. Secondary Outcome: Number of Participants With Symptomatic AEs Measured by Patient-reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: The PRO-CTCAE is a patient-reported outcome measure developed to evaluate symptomatic toxicity in participants on cancer clinical trials. It included symptomatic toxicities drawn from the CTCAE like blurred vision, chills, constipation, decreased appetite, fatigue, general pain, heart palpitations, mouth/throat sores, nausea, nosebleed, shortness of breath, vomiting and watery eyes. Items were scored individually on a 0 to 4 scale for severity, frequency and interference. Number of participants with symptomatic AEs (those who had a maximum post-Baseline rating greater than 0, example; 1, 2, 3, or 4) measured by PRO-CTCAE are presented.
Time Frame: Up to 186 weeks
Population: Full Safety Population. 3 participants out of 221 participants did not receive any study treatment and thus, were excluded from the Full Safety Population. only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 84 | 92 | 22
Participants
  Blurred Vision, n= 84,92,22 | 59 | 67 | 19
  Chills, n=43,42,13: number analyzed (Participants) | 43 | 42 | 13
  Chills, n=43,42,13 | 39 | 36 | 12
  Constipation, n=84,92, 22 | 42 | 47 | 17
  Decreased Appetite, n=84,92, 22 | 60 | 65 | 16
  Fatigue, n=84,92, 22 | 81 | 87 | 21
  General Pain, n= 79, 80, 20: number analyzed (Participants) | 79 | 80 | 20
  General Pain, n= 79, 80, 20 | 78 | 80 | 19
  Heart Palpitations, n=37, 37, 14: number analyzed (Participants) | 37 | 37 | 14
  Heart Palpitations, n=37, 37, 14 | 35 | 33 | 14
  Mouth/Throat Sores, n=84,92, 22 | 28 | 25 | 8
  Nausea, n=48, 52, 11: number analyzed (Participants) | 48 | 52 | 11
  Nausea, n=48, 52, 11 | 47 | 50 | 11
  Nosebleed, n=23, 33, 6: number analyzed (Participants) | 23 | 33 | 6
  Nosebleed, n=23, 33, 6 | 22 | 33 | 6
  Shortness Of Breath, n=84,92, 22 | 60 | 58 | 17
  Vomiting, n=21, 28, 6: number analyzed (Participants) | 21 | 28 | 6
  Vomiting, n=21, 28, 6 | 20 | 28 | 5
  Watery Eyes, n=84,92, 22 | 50 | 59 | 19

59. Secondary Outcome: Worst Change From Baseline in National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) Overall Composite Score
Description: The NEI-VFQ-25 consisted of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question to assess the impact of ocular toxicity on visual function. Items were coded to a 0 to 100 scale and averaged to calculate domains. Domain scores ranged from 0 to 100; higher scores are better. Therefore, increase in score means improvement. Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Data for worst-case post Baseline is presented.
Time Frame: Baseline (Day 1) and up to Week 186
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 83 | 92 | 22
Scores on a scale | -20.0 (22.60) | -19.6 (21.66) | -23.1 (23.82)

60. Secondary Outcome: Worst Change From Baseline in Ocular Surface Disease Index (OSDI) Total Score
Description: The OSDI is a 12-item questionnaire designed to assess both the frequency of dry eye symptoms and their impact on vision-related functioning. The total OSDI score was calculated as (sum of scores for all questions answered*100) divided by (total number of questions answered*4). Domain scores ranged from 0 to 100; lower scores are better. Therefore, decrease in score from Baseline means improvement. Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Data for worst-case post Baseline is presented.
Time Frame: Baseline (Day 1) and up to Week 186
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 83 | 92 | 22
Scores on a scale | 26.9 (29.61) | 28.2 (28.49) | 35.0 (29.02)

61. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30-item Core Module (EORTC QLQ-C30) Score
Description: The EORTC QLQ-C30 includes 30-items with single and multi-item scales. These included five functional scales (physical functioning [PF], role functioning [RF], cognitive functioning [CF], emotional functioning [EF] and social functioning [SF]), three symptom scales (fatigue, pain and nausea/vomiting [N/V]), a global health status (GHS)/ Quality-of-Life (QoL) scale, and six single items (constipation, diarrhoea, insomnia, dyspnoea, appetite loss [AL] and financial difficulties [FD]). Response options are 1 to 4. Scores were averaged and transformed to 0 to 100, a high score for functional scales/ GHS/QoL represent better functioning ability or health-related quality-of-life (HRQoL), whereas a high score for symptom scales/ single items represent significant symptomatology. Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Week 07, Week 13, Week 19, Week 25, Week 31, Week 37, Week 43, Week 61, Week 79, Week 97, Week 115, Week 133, Week 151, Week 169, and Week 186
Population: Full Analysis Population. Only those participants who were measured analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 97 | 99 | 25
Scores on a scale
  GHS/QoL,Week 07,n=48,47,17: number analyzed (Participants) | 48 | 47 | 17
  GHS/QoL,Week 07,n=48,47,17 | -0.7 (20.47) | -4.1 (18.54) | 1.5 (23.80)
  GHS/QoL,Week 13,n=29,29,16: number analyzed (Participants) | 29 | 29 | 16
  GHS/QoL,Week 13,n=29,29,16 | -3.2 (18.42) | 6.0 (16.50) | 1.0 (14.23)
  GHS/QoL,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  GHS/QoL,Week 19,n=19,27,10 | -2.2 (13.84) | 3.7 (20.19) | 0 (12.42)
  GHS/QoL,Week 25,n=20,23,7: number analyzed (Participants) | 20 | 23 | 7
  GHS/QoL,Week 25,n=20,23,7 | -4.6 (16.10) | -2.5 (20.94) | 7.1 (8.91)
  GHS/QoL,Week 31,n=15,18,7: number analyzed (Participants) | 15 | 18 | 7
  GHS/QoL,Week 31,n=15,18,7 | -2.2 (14.59) | 5.1 (20.44) | 2.4 (14.20)
  GHS/QoL,Week 37,n=15,13,5: number analyzed (Participants) | 15 | 13 | 5
  GHS/QoL,Week 37,n=15,13,5 | -1.7 (14.50) | 1.9 (21.29) | 11.7 (4.56)
  GHS/QoL,Week 43,n=15,14,4: number analyzed (Participants) | 15 | 14 | 4
  GHS/QoL,Week 43,n=15,14,4 | -4.4 (14.04) | 10.7 (15.82) | 12.5 (10.76)
  GHS/QoL,Week 61,n=11,11,3: number analyzed (Participants) | 11 | 11 | 3
  GHS/QoL,Week 61,n=11,11,3 | -3.8 (17.23) | -5.3 (13.58) | 0.0 (0.00)
  GHS/QoL,Week 79,n=3,2,1: number analyzed (Participants) | 3 | 2 | 1
  GHS/QoL,Week 79,n=3,2,1 | 2.8 (24.06) | 16.7 (23.57) | 16.7 (NA) — NA indicates SD could not be calculated for a single participant.
  GHS/QoL,Week 97,n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  GHS/QoL,Week 97,n=4,5,3 | 8.3 (11.79) | 1.7 (25.28) | 8.3 (0.00)
  GHS/QoL,Week 115,n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  GHS/QoL,Week 115,n=2,6,3 | -4.2 (17.68) | 1.4 (22.00) | 2.8 (4.81)
  GHS/QoL,Week 133,n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  GHS/QoL,Week 133,n=2,1,2 | -4.2 (17.68) | 33.3 (NA) — NA indicates SD could not be calculated for a single participant. | -8.3 (11.79)
  GHS/QoL,Week 151,n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  GHS/QoL,Week 151,n=0,2,0 |  | 8.3 (35.36) |
  GHS/QoL,Week 169,n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  GHS/QoL,Week 169,n=0,1,0 |  | 33.3 (NA) — NA indicates SD could not be calculated for a single participant. |
  GHS/QoL,Week 186n=41,46,17: number analyzed (Participants) | 41 | 46 | 17
  GHS/QoL,Week 186n=41,46,17 | -8.1 (19.50) | -11.6 (22.46) | -3.9 (15.34)
  PF,,Week 07,n=48,47,17: number analyzed (Participants) | 48 | 47 | 17
  PF,,Week 07,n=48,47,17 | 4.4 (15.70) | -1.0 (21.93) | -5.5 (24.18)
  PF,Week 13, n=29,29,16: number analyzed (Participants) | 29 | 29 | 16
  PF,Week 13, n=29,29,16 | 0.7 (14.62) | 4.1 (11.19) | -12.5 (23.84)
  PF,,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  PF,,Week 19,n=19,27,10 | 0.4 (13.78) | 6.2 (24.87) | -4.0 (14.81)
  PF,Week 25, n=20,23,7: number analyzed (Participants) | 20 | 23 | 7
  PF,Week 25, n=20,23,7 | 1.3 (12.16) | 5.5 (25.08) | -1.0 (14.62)
  PF,Week 31,n=15,18,7: number analyzed (Participants) | 15 | 18 | 7
  PF,Week 31,n=15,18,7 | -2.7 (8.66) | 9.3 (22.88) | 4.8 (10.69)
  PF, Week 37,n=15,13, 5: number analyzed (Participants) | 15 | 13 | 5
  PF, Week 37,n=15,13, 5 | 4.0 (11.76) | 15.4 (25.15) | 10.7 (18.62)
  PF, Week 43,n=15,14, 4: number analyzed (Participants) | 15 | 14 | 4
  PF, Week 43,n=15,14, 4 | 3.1 (11.23) | 14.8 (26.04) | 6.7 (27.22)
  PF, Week 61,n=11,11, 3: number analyzed (Participants) | 11 | 11 | 3
  PF, Week 61,n=11,11, 3 | 4.2 (12.39) | 9.7 (22.18) | 15.6 (3.85)
  PF, Week 79,n=3,2, 2: number analyzed (Participants) | 3 | 2 | 2
  PF, Week 79,n=3,2, 2 | 2.2 (3.85) | 10.0 (4.71) | 10.0 (4.71)
  PF, Week 97,n=4,5, 3: number analyzed (Participants) | 4 | 5 | 3
  PF, Week 97,n=4,5, 3 | 0.0 (9.43) | 0.0 (9.43) | -2.2 (23.41)
  PF, Week 115,n=2,6, 3: number analyzed (Participants) | 2 | 6 | 3
  PF, Week 115,n=2,6, 3 | 3.3 (4.71) | 4.4 (13.11) | 4.4 (10.18)
  PF, Week 133,n=2,1, 2: number analyzed (Participants) | 2 | 1 | 2
  PF, Week 133,n=2,1, 2 | 3.3 (4.71) | 13.3 (NA) — NA indicates SD could not be calculated for a single participant. | -6.7 (18.86)
  PF, Week 151,n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  PF, Week 151,n=0,2,0 |  | 0.0 (18.86) |
  PF, Week 169, n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  PF, Week 169, n=0,1,0 |  | 13.3 (NA) — NA indicates SD could not be calculated for a single participant. |
  PF, Week 186,n=41,46,17: number analyzed (Participants) | 41 | 46 | 17
  PF, Week 186,n=41,46,17 | -0.8 (21.20) | -6.2 (21.29) | -13.3 (24.38)
  RF,Week 07,n=48,47,17: number analyzed (Participants) | 48 | 47 | 17
  RF,Week 07,n=48,47,17 | 0.3 (33.24) | -6.0 (35.68) | -7.8 (25.08)
  RF,Week 13,n=29,29,16: number analyzed (Participants) | 29 | 29 | 16
  RF,Week 13,n=29,29,16 | 2.3 (33.55) | -0.6 (32.88) | -6.3 (30.96)
  RF,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  RF,Week 19,n=19,27,10 | -4.4 (31.35) | 1.9 (36.50) | -5.0 (23.64)
  RF,Week 25,n=20,23,7: number analyzed (Participants) | 20 | 23 | 7
  RF,Week 25,n=20,23,7 | 2.5 (32.57) | 0.0 (32.57) | 11.9 (32.93)
  RF,Week 31,n=15,18,7: number analyzed (Participants) | 15 | 18 | 7
  RF,Week 31,n=15,18,7 | 8.9 (24.29) | 3.7 (34.09) | 7.1 (21.21)
  RF,Week 37,n=15,13,5: number analyzed (Participants) | 15 | 13 | 5
  RF,Week 37,n=15,13,5 | 8.9 (29.46) | 3.8 (39.76) | 20.0 (27.39)
  RF,Week 43,n=15,14,4: number analyzed (Participants) | 15 | 14 | 4
  RF,Week 43,n=15,14,4 | 8.9 (30.12) | 11.9 (32.31) | 8.3 (21.52)
  RF,Week 61,n=11,11,3: number analyzed (Participants) | 11 | 11 | 3
  RF,Week 61,n=11,11,3 | 12.1 (36.58) | -3.0 (29.64) | 16.7 (16.67)
  RF,Week 79,n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  RF,Week 79,n=3,2,2 | 5.6 (34.69) | 8.3 (11.79) | 8.3 (35.36)
  RF,Week 97,n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  RF,Week 97,n=4,5,3 | -4.2 (43.83) | -6.7 (19.00) | 5.6 (34.69)
  RF,Week 115,n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  RF,Week 115,n=2,6,3 | 0.0 (47.14) | -5.6 (17.21) | 16.7 (44.10)
  RF,Week 133,n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  RF,Week 133,n=2,1,2 | 8.3 (35.36) | 16.7 (NA) — NA indicates SD could not be calculated for a single participant. | 25.0 (11.79)
  RF,Week 151,n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  RF,Week 151,n=0,2,0 |  | -16.7 (23.57) |
  RF,Week 169,n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  RF,Week 169,n=0,1,0 |  | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. |
  RF,Week 186,n=41,46,17: number analyzed (Participants) | 41 | 46 | 17
  RF,Week 186,n=41,46,17 | -0.4 (30.84) | -8.3 (33.66) | -16.7 (30.62)
  EF,Week 07,n=48,47,17: number analyzed (Participants) | 48 | 47 | 17
  EF,Week 07,n=48,47,17 | 1.4 (18.86) | 1.4 (27.10) | -4.4 (21.27)
  EF,Week 13,n=29,29,16: number analyzed (Participants) | 29 | 29 | 16
  EF,Week 13,n=29,29,16 | -2.0 (23.00) | -0.0 (25.00) | -9.4 (23.35)
  EF,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  EF,Week 19,n=19,27,10 | 0.4 (19.93) | 3.1 (20.30) | -1.7 (21.08)
  EF,Week 25, n=20, 23, 7: number analyzed (Participants) | 20 | 23 | 7
  EF,Week 25, n=20, 23, 7 | -4.6 (21.20) | 4.0 (20.39) | -2.4 (14.20)
  EF,Week 31, n=15,18, 7: number analyzed (Participants) | 15 | 18 | 7
  EF,Week 31, n=15,18, 7 | 2.2 (19.53) | 0.9 (25.06) | 1.2 (18.28)
  EF,Week 37, n=15,13, 5: number analyzed (Participants) | 15 | 13 | 5
  EF,Week 37, n=15,13, 5 | 1.7 (13.44) | 9.6 (23.29) | 13.3 (16.24)
  EF,Week 43, n=15,14, 4: number analyzed (Participants) | 15 | 14 | 4
  EF,Week 43, n=15,14, 4 | 0.0 (18.90) | 8.3 (27.74) | 4.2 (4.81)
  EF,Week 61, n=11,11, 3: number analyzed (Participants) | 11 | 11 | 3
  EF,Week 61, n=11,11, 3 | 6.8 (12.81) | -5.3 (16.36) | 19.4 (12.73)
  EF,Week 79, n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  EF,Week 79, n=3,2,2 | 2.8 (4.81) | 8.3 (11.79) | 16.7 (23.57)
  EF,Week 97, n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  EF,Week 97, n=4,5,3 | 2.1 (10.49) | 1.7 (25.95) | 8.3 (16.67)
  EF,Week 115, n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  EF,Week 115, n=2,6,3 | 0.0 (23.57) | -2.8 (11.39) | 11.1 (12.73)
  EF,Week 133, n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  EF,Week 133, n=2,1,2 | -4.2 (29.46) | 16.7 (NA) — NA indicates SD could not be calculated for a single participant. | 8.3 (23.57)
  EF,Week 151, n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  EF,Week 151, n=0,2,0 |  | 4.2 (29.46) |
  EF,Week 169, n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  EF,Week 169, n=0,1,0 |  | 16.7 (NA) — NA indicates SD could not be calculated for a single participant. |
  EF,Week 186, n=41,46,17: number analyzed (Participants) | 41 | 46 | 17
  EF,Week 186, n=41,46,17 | -6.7 (24.45) | -6.2 (21.04) | -10.8 (17.37)
  CF,Week 07,n=48,47,17: number analyzed (Participants) | 48 | 47 | 17
  CF,Week 07,n=48,47,17 | 4.5 (20.55) | -2.1 (21.03) | -1.0 (20.81)
  CF,Week 13,n=29,29,16: number analyzed (Participants) | 29 | 29 | 16
  CF,Week 13,n=29,29,16 | 2.3 (23.45) | -1.1 (15.39) | -15.6 (27.53)
  CF,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  CF,Week 19,n=19,27,10 | -1.8 (26.58) | -0.6 (22.87) | -6.7 (21.08)
  CF,Week 25, n=20, 23, 7: number analyzed (Participants) | 20 | 23 | 7
  CF,Week 25, n=20, 23, 7 | -1.7 (27.52) | 1.4 (21.27) | -11.9 (18.54)
  CF,Week 31, n=15,18, 7: number analyzed (Participants) | 15 | 18 | 7
  CF,Week 31, n=15,18, 7 | 6.7 (23.40) | -3.7 (19.43) | -4.8 (12.60)
  CF,Week 37, n=15,13, 5: number analyzed (Participants) | 15 | 13 | 5
  CF,Week 37, n=15,13, 5 | 3.3 (22.00) | 3.8 (13.87) | 3.3 (13.94)
  CF,Week 43, n=15,14, 4: number analyzed (Participants) | 15 | 14 | 4
  CF,Week 43, n=15,14, 4 | 2.2 (24.29) | 1.2 (10.26) | -4.2 (8.33)
  CF,Week 61, n=11,11, 3: number analyzed (Participants) | 11 | 11 | 3
  CF,Week 61, n=11,11, 3 | 10.6 (27.15) | -1.5 (15.73) | 5.6 (9.62)
  CF,Week 79, n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  CF,Week 79, n=3,2,2 | 11.1 (19.25) | -25.0 (35.36) | 8.3 (11.79)
  CF,Week 97, n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  CF,Week 97, n=4,5,3 | -4.2 (25.00) | -16.7 (33.33) | 0.0 (16.67)
  CF,Week 115, n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  CF,Week 115, n=2,6,3 | 0.0 (23.57) | -0.0 (18.26) | 11.1 (9.62)
  CF,Week 133, n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  CF,Week 133, n=2,1,2 | -8.3 (35.36) | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. | 8.3 (11.79)
  CF,Week 151, n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  CF,Week 151, n=0,2,0 |  | -16.7 (23.57) |
  CF,Week 169, n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  CF,Week 169, n=0,1,0 |  | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. |
  CF,Week 186, n=41,46,17: number analyzed (Participants) | 41 | 46 | 17
  CF,Week 186, n=41,46,17 | -3.3 (25.88) | -11.2 (26.07) | -9.8 (13.25)
  SF,Week 07,n=48,47,17: number analyzed (Participants) | 48 | 47 | 17
  SF,Week 07,n=48,47,17 | 3.8 (29.02) | 1.1 (32.49) | -1.0 (33.58)
  SF,Week 13,n=29,29,16: number analyzed (Participants) | 29 | 29 | 16
  SF,Week 13,n=29,29,16 | -4.0 (28.75) | 1.7 (28.64) | -7.3 (31.01)
  SF,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  SF,Week 19,n=19,27,10 | -6.1 (28.44) | 5.6 (28.50) | -6.7 (28.54)
  SF,Week 25, n=20, 23, 7: number analyzed (Participants) | 20 | 23 | 7
  SF,Week 25, n=20, 23, 7 | -6.7 (26.71) | 13.8 (22.84) | 2.4 (32.53)
  SF,Week 31, n=15,18, 7: number analyzed (Participants) | 15 | 18 | 7
  SF,Week 31, n=15,18, 7 | 2.2 (16.51) | 15.7 (31.56) | 2.4 (24.40)
  SF,Week 37, n=15,13, 5: number analyzed (Participants) | 15 | 13 | 5
  SF,Week 37, n=15,13, 5 | 2.2 (21.70) | 16.7 (29.66) | 20.0 (21.73)
  SF,Week 43, n=15,14, 4: number analyzed (Participants) | 15 | 14 | 4
  SF,Week 43, n=15,14, 4 | -1.1 (17.21) | 20.2 (30.08) | 16.7 (23.57)
  SF,Week 61, n=11,11, 3: number analyzed (Participants) | 11 | 11 | 3
  SF,Week 61, n=11,11, 3 | 7.6 (32.80) | -1.5 (17.41) | 33.3 (16.67)
  SF,Week 79, n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  SF,Week 79, n=3,2,2 | 5.6 (19.25) | 8.3 (35.36) | 25.0 (35.36)
  SF,Week 97, n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  SF,Week 97, n=4,5,3 | -4.2 (43.83) | 16.7 (20.41) | 33.3 (16.67)
  SF,Week 115, n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  SF,Week 115, n=2,6,3 | 16.7 (23.57) | 2.8 (24.53) | 27.8 (25.46)
  SF,Week 133, n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  SF,Week 133, n=2,1,2 | 16.7 (23.57) | 33.3 (NA) — NA indicates SD could not be calculated for a single participant. | 41.7 (11.79)
  SF,Week 151, n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  SF,Week 151, n=0,2,0 |  | 16.7 (23.57) |
  SF,Week 169, n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  SF,Week 169, n=0,1,0 |  | 33.3 (NA) — NA indicates SD could not be calculated for a single participant. |
  SF,Week 186, n=41,46,17: number analyzed (Participants) | 41 | 46 | 17
  SF,Week 186, n=41,46,17 | -4.1 (26.56) | -10.1 (25.93) | -8.8 (31.80)
  Fatigue,Week 07,n=48,47,17: number analyzed (Participants) | 48 | 47 | 17
  Fatigue,Week 07,n=48,47,17 | -3.7 (21.90) | -0.5 (23.74) | -5.2 (20.83)
  Fatigue,Week 13,n=29,29,16: number analyzed (Participants) | 29 | 29 | 16
  Fatigue,Week 13,n=29,29,16 | -7.7 (23.78) | -7.7 (19.27) | -1.4 (24.97)
  Fatigue,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  Fatigue,Week 19,n=19,27,10 | -0.6 (22.67) | -2.9 (22.77) | -11.1 (15.71)
  Fatigue,Week 25, n=20, 23, 7: number analyzed (Participants) | 20 | 23 | 7
  Fatigue,Week 25, n=20, 23, 7 | 3.3 (23.67) | -2.4 (21.70) | -11.1 (16.97)
  Fatigue,Week 31, n=15,18, 7: number analyzed (Participants) | 15 | 18 | 7
  Fatigue,Week 31, n=15,18, 7 | -0.7 (21.61) | -11.7 (22.05) | -12.7 (18.62)
  Fatigue,Week 37, n=15,13, 5: number analyzed (Participants) | 15 | 13 | 5
  Fatigue,Week 37, n=15,13, 5 | -9.6 (18.24) | -13.7 (24.07) | -20.0 (14.49)
  Fatigue,Week 43, n=15,14, 4: number analyzed (Participants) | 15 | 14 | 4
  Fatigue,Week 43, n=15,14, 4 | -12.6 (17.25) | -10.3 (32.16) | -22.2 (12.83)
  Fatigue,Week 61, n=11,11, 3: number analyzed (Participants) | 11 | 11 | 3
  Fatigue,Week 61, n=11,11, 3 | -12.1 (24.07) | 3.0 (22.82) | -11.1 (0.00)
  Fatigue,Week 79, n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  Fatigue,Week 79, n=3,2,2 | -22.2 (11.11) | -16.7 (7.86) | 5.6 (23.57)
  Fatigue,Week 97, n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  Fatigue,Week 97, n=4,5,3 | -5.6 (26.45) | 6.7 (20.18) | -25.9 (23.13)
  Fatigue,Week 115, n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  Fatigue,Week 115, n=2,6,3 | -16.7 (23.57) | -3.7 (15.18) | -18.5 (23.13)
  Fatigue,Week 133, n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  Fatigue,Week 133, n=2,1,2 | -5.6 (39.28) | -22.2 (NA) — NA indicates SD could not be calculated for a single participant. | -22.2 (15.71)
  Fatigue,Week 151, n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  Fatigue,Week 151, n=0,2,0 |  | 16.7 (23.57) |
  Fatigue,Week 169, n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  Fatigue,Week 169, n=0,1,0 |  | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. |
  Fatigue,Week 186, n=41,46,17: number analyzed (Participants) | 41 | 46 | 17
  Fatigue,Week 186, n=41,46,17 | -1.6 (23.12) | 4.1 (23.35) | 6.5 (22.93)
  N/V,Week 07,n=48,47,17: number analyzed (Participants) | 48 | 47 | 17
  N/V,Week 07,n=48,47,17 | 2.4 (14.17) | 4.3 (17.88) | 2.0 (14.29)
  N/V,Week 13,n=29,29,16: number analyzed (Participants) | 29 | 29 | 16
  N/V,Week 13,n=29,29,16 | 2.3 (13.16) | 1.1 (9.89) | 7.3 (25.80)
  N/V,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  N/V,Week 19,n=19,27,10 | -1.8 (15.61) | -1.2 (15.96) | 1.7 (5.27)
  N/V,Week 25,n=20,23,7: number analyzed (Participants) | 20 | 23 | 7
  N/V,Week 25,n=20,23,7 | 5.0 (12.21) | -0.7 (12.79) | -4.8 (12.60)
  N/V,Week 31,n=15,18,7: number analyzed (Participants) | 15 | 18 | 7
  N/V,Week 31,n=15,18,7 | -3.3 (6.90) | 1.9 (7.86) | -2.4 (15.00)
  N/V,Week 37,n=15,13, 5: number analyzed (Participants) | 15 | 13 | 5
  N/V,Week 37,n=15,13, 5 | -6.7 (16.43) | 2.6 (11.48) | 0.0 (0.00)
  N/V,Week 43,n=15,14,4: number analyzed (Participants) | 15 | 14 | 4
  N/V,Week 43,n=15,14,4 | -7.8 (15.26) | 1.2 (7.91) | -8.3 (16.67)
  N/V,Week 61, n=11,11,3: number analyzed (Participants) | 11 | 11 | 3
  N/V,Week 61, n=11,11,3 | -4.5 (10.78) | 4.5 (7.78) | 0.0 (16.67)
  N/V,Week 79, n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  N/V,Week 79, n=3,2,2 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  N/V,Week 97, n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  N/V,Week 97, n=4,5,3 | 0.0 (0.00) | 0.0 (0.00) | -11.1 (19.25)
  N/V,Week 115, n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  N/V,Week 115, n=2,6,3 | 0.0 (0.00) | 0.0 (0.00) | -16.7 (16.67)
  N/V,Week 133, n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  N/V,Week 133, n=2,1,2 | 0.0 (0.00) | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. | -25.0 (11.79)
  N/V, Week 151, n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  N/V, Week 151, n=0,2,0 |  | 0.0 (0.00) |
  N/V, Week 169, n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  N/V, Week 169, n=0,1,0 |  | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. |
  N/V, Week 186, n=41,46,17: number analyzed (Participants) | 41 | 46 | 17
  N/V, Week 186, n=41,46,17 | 5.7 (24.04) | 3.3 (18.47) | 1.0 (21.63)
  Pain,Week 07,n=48,47,17: number analyzed (Participants) | 48 | 47 | 17
  Pain,Week 07,n=48,47,17 | -3.1 (28.69) | -1.1 (28.32) | 8.8 (28.33)
  Pain,Week 13,n=29,28,16: number analyzed (Participants) | 29 | 28 | 16
  Pain,Week 13,n=29,28,16 | -4.0 (26.97) | -2.3 (25.48) | 5.2 (27.02)
  Pain,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  Pain,Week 19,n=19,27,10 | 4.4 (19.12) | -8.6 (31.14) | 1.7 (30.88)
  Pain,Week 25,n=20,23,7: number analyzed (Participants) | 20 | 23 | 7
  Pain,Week 25,n=20,23,7 | 2.5 (18.16) | -1.4 (24.57) | -0.0 (28.87)
  Pain,Week 31,n=15,18,7: number analyzed (Participants) | 15 | 18 | 7
  Pain,Week 31,n=15,18,7 | 4.4 (19.38) | -0.9 (23.90) | 2.4 (35.26)
  Pain,Week 37,n=15,13,5: number analyzed (Participants) | 15 | 13 | 5
  Pain,Week 37,n=15,13,5 | -2.2 (21.70) | -10.3 (24.09) | -3.3 (24.72)
  Pain,Week 43,n=15,14,4: number analyzed (Participants) | 15 | 14 | 4
  Pain,Week 43,n=15,14,4 | -2.2 (15.26) | -8.3 (24.24) | 4.2 (36.96)
  Pain,Week 61,n=11,11,3: number analyzed (Participants) | 11 | 11 | 3
  Pain,Week 61,n=11,11,3 | -10.6 (18.67) | -0.0 (21.08) | -5.6 (34.69)
  Pain,Week 79,n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  Pain,Week 79,n=3,2,2 | -16.7 (16.67) | 0.0 (23.57) | 8.3 (58.93)
  Pain,Week 97,n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  Pain,Week 97,n=4,5,3 | -4.2 (20.97) | 26.7 (22.36) | -0.0 (44.10)
  Pain,Week 115,n=2,6, 3: number analyzed (Participants) | 2 | 6 | 3
  Pain,Week 115,n=2,6, 3 | 0.0 (0.00) | 8.3 (27.39) | 5.6 (53.58)
  Pain,Week 133,n=2,1, 2: number analyzed (Participants) | 2 | 1 | 2
  Pain,Week 133,n=2,1, 2 | 0.0 (0.00) | 16.7 (NA) — NA indicates SD could not be calculated for a single participant. | 16.7 (70.71)
  Pain,Week 151,n=0,2, 0: number analyzed (Participants) | 0 | 2 | 0
  Pain,Week 151,n=0,2, 0 |  | 33.3 (23.57) |
  Pain,Week 169,n=0,1, 0: number analyzed (Participants) | 0 | 1 | 0
  Pain,Week 169,n=0,1, 0 |  | 16.7 |
  Pain,Week 186,n=41,46, 17: number analyzed (Participants) | 41 | 46 | 17
  Pain,Week 186,n=41,46, 17 | 1.6 (27.59) | 1.4 (25.29) | 16.7 (31.73)
  Dyspnoea,Week 07,n=48,47,17: number analyzed (Participants) | 48 | 47 | 17
  Dyspnoea,Week 07,n=48,47,17 | -2.1 (22.18) | 2.1 (14.59) | -7.8 (18.74)
  Dyspnoea,Week 13,n=29,29,16: number analyzed (Participants) | 29 | 29 | 16
  Dyspnoea,Week 13,n=29,29,16 | -1.1 (18.86) | 1.1 (22.68) | 2.1 (30.96)
  Dyspnoea,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  Dyspnoea,Week 19,n=19,27,10 | -5.3 (20.07) | 3.7 (25.04) | -16.7 (28.33)
  Dyspnoea,Week 25,n=20,23,7: number analyzed (Participants) | 20 | 23 | 7
  Dyspnoea,Week 25,n=20,23,7 | -1.7 (20.16) | 4.3 (18.27) | 0.0 (27.22)
  Dyspnoea,Week 31,n=15, 18, 7: number analyzed (Participants) | 15 | 18 | 7
  Dyspnoea,Week 31,n=15, 18, 7 | -6.7 (18.69) | 0.0 (16.17) | -9.5 (16.27)
  Dyspnoea,Week 37,n=15, 13, 5: number analyzed (Participants) | 15 | 13 | 5
  Dyspnoea,Week 37,n=15, 13, 5 | -8.9 (19.79) | 12.8 (16.88) | -26.7 (27.89)
  Dyspnoea,Week 43,n=15, 14, 4: number analyzed (Participants) | 15 | 14 | 4
  Dyspnoea,Week 43,n=15, 14, 4 | -6.7 (22.54) | 2.4 (15.82) | -25.0 (31.91)
  Dyspnoea,Week 61,n=11,11,3: number analyzed (Participants) | 11 | 11 | 3
  Dyspnoea,Week 61,n=11,11,3 | 0.0 (21.08) | 3.0 (17.98) | -33.3 (33.33)
  Dyspnoea,Week 79,n=3, 2,2: number analyzed (Participants) | 3 | 2 | 2
  Dyspnoea,Week 79,n=3, 2,2 | 0.0 (0.00) | 0.0 (0.00) | -33.3 (47.14)
  Dyspnoea,Week 97,n=4, 5,3: number analyzed (Participants) | 4 | 5 | 3
  Dyspnoea,Week 97,n=4, 5,3 | 16.7 (19.25) | 0.0 (23.57) | -22.2 (38.49)
  Dyspnoea,Week 115,n=2, 6,3: number analyzed (Participants) | 2 | 6 | 3
  Dyspnoea,Week 115,n=2, 6,3 | 0.0 (0.00) | 5.6 (13.61) | -33.3 (33.33)
  Dyspnoea,Week 133,n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  Dyspnoea,Week 133,n=2,1,2 | 0.0 (0.00) | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. | -16.7 (23.57)
  Dyspnoea,Week 151,n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  Dyspnoea,Week 151,n=0,2,0 |  | 0.0 (0.00) |
  Dyspnoea,Week 169,n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  Dyspnoea,Week 169,n=0,1,0 |  | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. |
  Dyspnoea,Week 186,n=41, 46,17: number analyzed (Participants) | 41 | 46 | 17
  Dyspnoea,Week 186,n=41, 46,17 | 0.0 (19.72) | 12.3 (24.70) | -9.8 (25.72)
  Insomnia,Week 07,n=48, 47, 17: number analyzed (Participants) | 48 | 47 | 17
  Insomnia,Week 07,n=48, 47, 17 | -6.2 (29.70) | -2.8 (26.77) | -0.0 (23.57)
  Insomnia,Week 13,n=29,29,16: number analyzed (Participants) | 29 | 29 | 16
  Insomnia,Week 13,n=29,29,16 | 0.0 (26.73) | -1.1 (25.95) | -0.0 (34.43)
  Insomnia,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  Insomnia,Week 19,n=19,27,10 | -8.8 (24.45) | -4.9 (28.80) | -13.3 (35.83)
  Insomnia,Week 25,n=20,23,7: number analyzed (Participants) | 20 | 23 | 7
  Insomnia,Week 25,n=20,23,7 | -5.0 (32.94) | -7.2 (22.38) | 0.0 (33.33)
  Insomnia,Week 31,n=15,18,7: number analyzed (Participants) | 15 | 18 | 7
  Insomnia,Week 31,n=15,18,7 | -17.8 (27.79) | -9.3 (33.93) | 4.8 (40.50)
  Insomnia,Week 37,n=15,13,5: number analyzed (Participants) | 15 | 13 | 5
  Insomnia,Week 37,n=15,13,5 | -15.6 (33.01) | -10.3 (16.01) | -13.3 (38.01)
  Insomnia,Week 43,n=15,14,4: number analyzed (Participants) | 15 | 14 | 4
  Insomnia,Week 43,n=15,14,4 | -15.6 (30.52) | -4.8 (22.10) | -0.0 (47.14)
  Insomnia,Week 61,n=11,11,3: number analyzed (Participants) | 11 | 11 | 3
  Insomnia,Week 61,n=11,11,3 | -9.1 (15.57) | -9.1 (21.56) | -11.1 (19.25)
  Insomnia,Week 79,n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  Insomnia,Week 79,n=3,2,2 | 0.0 (33.33) | 16.7 (23.57) | -33.3 (47.14)
  Insomnia,Week 97,n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  Insomnia,Week 97,n=4,5,3 | -25.0 (31.91) | -6.7 (14.91) | -44.4 (38.49)
  Insomnia,Week 115,n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  Insomnia,Week 115,n=2,6,3 | -33.3 (47.14) | 5.6 (25.09) | -33.3 (33.33)
  Insomnia,Week 133,n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  Insomnia,Week 133,n=2,1,2 | -16.7 (70.71) | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. | -66.7 (0.00)
  Insomnia,Week 151,n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  Insomnia,Week 151,n=0,2,0 |  | 0.0 (0.00) |
  Insomnia,Week 169,n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  Insomnia,Week 169,n=0,1,0 |  | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. |
  Insomnia,Week 186,n=41,46,17: number analyzed (Participants) | 41 | 46 | 17
  Insomnia,Week 186,n=41,46,17 | 2.4 (33.66) | -2.9 (32.07) | 2.0 (29.98)
  AL,Week 07,n=48,47,17: number analyzed (Participants) | 48 | 47 | 17
  AL,Week 07,n=48,47,17 | 4.9 (24.78) | 2.1 (29.00) | 2.0 (27.56)
  AL,Week 13,n=29,29,16: number analyzed (Participants) | 29 | 29 | 16
  AL,Week 13,n=29,29,16 | 8.0 (29.08) | -2.3 (25.09) | 12.5 (26.87)
  AL,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  AL,Week 19,n=19,27,10 | 0.0 (24.85) | -0.0 (38.12) | -3.3 (10.54)
  AL,Week 25,n=20, 23, 7: number analyzed (Participants) | 20 | 23 | 7
  AL,Week 25,n=20, 23, 7 | 6.7 (31.72) | -5.8 (21.68) | -9.5 (16.27)
  AL,Week 31,n=15,18, 7: number analyzed (Participants) | 15 | 18 | 7
  AL,Week 31,n=15,18, 7 | -8.9 (15.26) | 0.0 (19.80) | -4.8 (23.00)
  AL,Week 37,n=15,13,5: number analyzed (Participants) | 15 | 13 | 5
  AL,Week 37,n=15,13,5 | -4.4 (17.21) | -5.1 (22.96) | -20.0 (18.26)
  AL,Week 43,n=15,14,4: number analyzed (Participants) | 15 | 14 | 4
  AL,Week 43,n=15,14,4 | -4.4 (17.21) | -9.5 (24.21) | -25.0 (16.67)
  AL,Week 61,n=11,11,3: number analyzed (Participants) | 11 | 11 | 3
  AL,Week 61,n=11,11,3 | -6.1 (20.10) | 0.0 (36.51) | 11.1 (19.25)
  AL,Week 79,n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  AL,Week 79,n=3,2,2 | -33.3 (0.00) | 16.7 (23.57) | 16.7 (23.57)
  AL,Week 97,n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  AL,Week 97,n=4,5,3 | -8.3 (16.67) | 13.3 (18.26) | 0.0 (33.33)
  AL,Week 115,n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  AL,Week 115,n=2,6,3 | 0.0 (0.00) | 0.0 (21.08) | 0.0 (33.33)
  AL,Week 133,n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  AL,Week 133,n=2,1,2 | 0.0 (0.00) | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. | -16.7 (23.57)
  AL,Week 151,n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  AL,Week 151,n=0,2,0 |  | 33.3 (47.14) |
  AL,Week 169,n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  AL,Week 169,n=0,1,0 |  | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. |
  AL,Week 186,n=41,46,17: number analyzed (Participants) | 41 | 46 | 17
  AL,Week 186,n=41,46,17 | 5.7 (24.61) | -0.0 (32.96) | 2.0 (21.96)
  Constipation,Week 07,n=48,47,17: number analyzed (Participants) | 48 | 47 | 17
  Constipation,Week 07,n=48,47,17 | 1.4 (22.76) | -2.1 (17.59) | -7.8 (25.08)
  Constipation,Week 13,n=29,29,16: number analyzed (Participants) | 29 | 29 | 16
  Constipation,Week 13,n=29,29,16 | 0.0 (25.20) | -5.7 (17.97) | 8.3 (31.03)
  Constipation,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  Constipation,Week 19,n=19,27,10 | -7.0 (21.02) | 1.2 (17.25) | -3.3 (18.92)
  Constipation,Week 25,n=20,23,7: number analyzed (Participants) | 20 | 23 | 7
  Constipation,Week 25,n=20,23,7 | -3.3 (14.91) | -1.4 (18.74) | -14.3 (32.53)
  Constipation,Week 31,n=15,18,7: number analyzed (Participants) | 15 | 18 | 7
  Constipation,Week 31,n=15,18,7 | -4.4 (11.73) | -3.7 (15.71) | -19.0 (26.23)
  Constipation,Week 37,n=15,13,5: number analyzed (Participants) | 15 | 13 | 5
  Constipation,Week 37,n=15,13,5 | 2.2 (23.46) | -5.1 (22.96) | -20.0 (38.01)
  Constipation,Week 43,n=15,14,4: number analyzed (Participants) | 15 | 14 | 4
  Constipation,Week 43,n=15,14,4 | -4.4 (17.21) | -2.4 (20.52) | -16.7 (43.03)
  Constipation,Week 61,n=11,11,3: number analyzed (Participants) | 11 | 11 | 3
  Constipation,Week 61,n=11,11,3 | 0.0 (14.91) | -9.1 (30.15) | -11.1 (38.49)
  Constipation,Week 79,n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  Constipation,Week 79,n=3,2,2 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (47.14)
  Constipation,Week 97,n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  Constipation,Week 97,n=4,5,3 | 0.0 (0.00) | 0.0 (0.00) | -22.2 (50.92)
  Constipation,Week 115,n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  Constipation,Week 115,n=2,6,3 | 0.0 (0.00) | -5.6 (13.61) | -22.2 (50.92)
  Constipation,Week 133,n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  Constipation,Week 133,n=2,1,2 | 0.0 (0.00) | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. | -50.0 (23.57)
  Constipation,Week 151,n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  Constipation,Week 151,n=0,2,0 |  | 0.0 (0.00) |
  Constipation,Week 169,n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  Constipation,Week 169,n=0,1,0 |  | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. |
  Constipation,Week 186,n=41,46,17: number analyzed (Participants) | 41 | 46 | 17
  Constipation,Week 186,n=41,46,17 | 5.7 (20.95) | 3.6 (20.16) | 3.9 (33.09)
  Diarrhoea,Week 07,n=48,47,17: number analyzed (Participants) | 48 | 47 | 17
  Diarrhoea,Week 07,n=48,47,17 | -2.8 (26.48) | -0.0 (28.66) | -2.0 (24.92)
  Diarrhoea,Week 13,n=29,29,16: number analyzed (Participants) | 29 | 29 | 16
  Diarrhoea,Week 13,n=29,29,16 | 0.0 (25.20) | -6.9 (18.64) | 4.2 (31.91)
  Diarrhoea,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  Diarrhoea,Week 19,n=19,27,10 | 1.8 (26.00) | -2.5 (24.33) | -3.3 (18.92)
  Diarrhoea,Week 25,n=20,23,7: number analyzed (Participants) | 20 | 23 | 7
  Diarrhoea,Week 25,n=20,23,7 | 3.3 (28.41) | -7.2 (33.27) | -19.0 (17.82)
  Diarrhoea,Week 31,n=15,18,7: number analyzed (Participants) | 15 | 18 | 7
  Diarrhoea,Week 31,n=15,18,7 | -2.2 (23.46) | -3.7 (34.09) | -4.8 (29.99)
  Diarrhoea,Week 37,n=15,13,5: number analyzed (Participants) | 15 | 13 | 5
  Diarrhoea,Week 37,n=15,13,5 | -2.2 (23.46) | 2.6 (28.74) | -20.0 (18.26)
  Diarrhoea,Week 43,n=15,14,4: number analyzed (Participants) | 15 | 14 | 4
  Diarrhoea,Week 43,n=15,14,4 | -4.4 (21.33) | 14.3 (28.39) | -16.7 (19.25)
  Diarrhoea,Week 61,n=11,11,3: number analyzed (Participants) | 11 | 11 | 3
  Diarrhoea,Week 61,n=11,11,3 | 0.0 (21.08) | 15.2 (31.14) | 0.0 (33.33)
  Diarrhoea,Week 79,n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  Diarrhoea,Week 79,n=3,2,2 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (47.14)
  Diarrhoea,Week 97,n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  Diarrhoea,Week 97,n=4,5,3 | -8.3 (16.67) | 0.0 (0.00) | -22.2 (19.25)
  Diarrhoea,Week 115,n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  Diarrhoea,Week 115,n=2,6,3 | 0.0 (0.00) | 0.0 (0.00) | -22.2 (19.25)
  Diarrhoea,Week 133,n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  Diarrhoea,Week 133,n=2,1,2 | 0.0 (0.00) | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. | -33.3 (0.00)
  Diarrhoea,Week 151,n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  Diarrhoea,Week 151,n=0,2,0 |  | 0.0 (0.00) |
  Diarrhoea,Week 169,n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  Diarrhoea,Week 169,n=0,1,0 |  | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. |
  Diarrhoea,Week 186,n=41,46,17: number analyzed (Participants) | 41 | 46 | 17
  Diarrhoea,Week 186,n=41,46,17 | -0.8 (21.72) | -5.1 (28.08) | 0.0 (35.36)
  FD,Week 07,n=48,47,17: number analyzed (Participants) | 48 | 47 | 17
  FD,Week 07,n=48,47,17 | -4.9 (25.72) | 2.8 (24.90) | 0.0 (16.67)
  FD,Week 13,n=29,29,16: number analyzed (Participants) | 29 | 29 | 16
  FD,Week 13,n=29,29,16 | -4.6 (23.10) | 4.6 (19.36) | 10.4 (20.07)
  FD,Week 19,n=19,27,10: number analyzed (Participants) | 19 | 27 | 10
  FD,Week 19,n=19,27,10 | -7.0 (21.02) | 3.7 (26.69) | 10.0 (22.50)
  FD,Week 25,n=20,23,7: number analyzed (Participants) | 20 | 23 | 7
  FD,Week 25,n=20,23,7 | -3.3 (26.27) | -1.4 (15.82) | 0.0 (19.25)
  FD,Week 31,n=15,18, 7: number analyzed (Participants) | 15 | 18 | 7
  FD,Week 31,n=15,18, 7 | -6.7 (22.54) | -1.9 (17.98) | 4.8 (23.00)
  FD,Week 37,n=15,13,5: number analyzed (Participants) | 15 | 13 | 5
  FD,Week 37,n=15,13,5 | -2.2 (23.46) | -2.6 (16.45) | 6.7 (14.91)
  FD,Week 43,n=15,14,4: number analyzed (Participants) | 15 | 14 | 4
  FD,Week 43,n=15,14,4 | -6.7 (18.69) | 0.0 (22.65) | 8.3 (31.91)
  FD,Week 61,n=11,11,3: number analyzed (Participants) | 11 | 11 | 3
  FD,Week 61,n=11,11,3 | -12.1 (37.34) | 6.1 (29.13) | 11.1 (19.25)
  FD,Week 79,n=3,2,1: number analyzed (Participants) | 3 | 2 | 1
  FD,Week 79,n=3,2,1 | 0.0 (0.00) | -16.7 (23.57) | 0.0 (NA) — NA indicates SD could not be calculated for a single participant.
  FD,Week 97,n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  FD,Week 97,n=4,5,3 | -25.0 (31.91) | 0.0 (23.57) | -11.1 (19.25)
  FD,Week 115,n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  FD,Week 115,n=2,6,3 | 0.0 (0.00) | 22.2 (50.18) | -11.1 (19.25)
  FD,Week 133,n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  FD,Week 133,n=2,1,2 | -50.0 (23.57) | -33.3 (NA) — NA indicates SD could not be calculated for a single participant. | -16.7 (23.57)
  FD,Week 151,n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  FD,Week 151,n=0,2,0 |  | -33.3 (0.00) |
  FD,Week 169,n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  FD,Week 169,n=0,1,0 |  | -33.3 (NA) — NA indicates SD could not be calculated for a single participant. |
  FD,Week 186,n=41,46,17: number analyzed (Participants) | 41 | 46 | 17
  FD,Week 186,n=41,46,17 | -1.6 (24.67) | 12.3 (25.68) | 5.9 (21.20)

62. Secondary Outcome: Change From Baseline in EORTC QLQ 20-item Multiple Myeloma Module (MY20) Score
Description: The EORTC QLQ-MY20 is a supplement to the QLQ-C30 instrument used in participants with multiple myeloma. The module comprised of 20 questions that addressed four myeloma-specific HRQoL domains: disease symptoms (DS), side effects of treatment (SET), future perspective (FP) and body image (BI). Responses are 1 to 4. Scores were averaged and scales were transformed to 0 to 100 scale. A high score for disease symptoms and side effects of treatment represented a high level of symptomatology or problems, whereas a high score for future perspective and body image represented better outcomes. Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: as for outcome 61
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized)
Number analyzed (Participants) | 97 | 99 | 25
Scores on a scale
  FP,Week 07,n=47,45,16: number analyzed (Participants) | 47 | 45 | 16
  FP,Week 07,n=47,45,16 | 2.8 (25.11) | 4.2 (29.99) | 8.3 (24.51)
  FP,Week 13,n=28,28,15: number analyzed (Participants) | 28 | 28 | 15
  FP,Week 13,n=28,28,15 | -2.0 (24.39) | 8.3 (22.55) | -2.2 (27.28)
  FP,Week 19,n=18,25,10: number analyzed (Participants) | 18 | 25 | 10
  FP,Week 19,n=18,25,10 | 3.7 (22.87) | 10.7 (20.91) | 3.3 (27.24)
  FP,Week 25,n=19,23,7: number analyzed (Participants) | 19 | 23 | 7
  FP,Week 25,n=19,23,7 | 2.3 (27.11) | 13.5 (29.39) | 4.8 (31.98)
  FP,Week 31,n=14,18,7: number analyzed (Participants) | 14 | 18 | 7
  FP,Week 31,n=14,18,7 | 7.1 (18.80) | 19.1 (24.93) | 7.9 (27.00)
  FP,Week 37,n=14,13,5: number analyzed (Participants) | 14 | 13 | 5
  FP,Week 37,n=14,13,5 | 6.3 (17.28) | 29.1 (22.47) | 11.1 (31.43)
  FP,Week 43,n=15,13,4: number analyzed (Participants) | 15 | 13 | 4
  FP,Week 43,n=15,13,4 | 8.1 (21.19) | 29.9 (26.98) | 8.3 (5.56)
  FP,Week 61,n=11,11,3: number analyzed (Participants) | 11 | 11 | 3
  FP,Week 61,n=11,11,3 | 10.1 (18.89) | 4.0 (20.65) | 25.9 (54.81)
  FP,Week 79,n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  FP,Week 79,n=3,2,2 | -7.4 (6.42) | 33.3 (31.43) | 38.9 (39.28)
  FP,Week 97,n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  FP,Week 97,n=4,5,3 | 5.6 (14.34) | 17.8 (39.75) | 22.2 (40.06)
  FP,Week 115,n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  FP,Week 115,n=2,6,3 | 11.1 (15.71) | 16.7 (25.09) | 33.3 (58.79)
  FP,Week 133,n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  FP,Week 133,n=2,1,2 | 27.8 (7.86) | 55.6 (NA) — NA indicates SD could not be calculated for a single participant. | 38.9 (55.00)
  FP,Week 151,n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  FP,Week 151,n=0,2,0 |  | 44.4 (15.71) |
  FP,Week 169,n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  FP,Week 169,n=0,1,0 |  | 55.6 (NA) — NA indicates SD could not be calculated for a single participant. |
  FP,Week 186,n=39,46,16: number analyzed (Participants) | 39 | 46 | 16
  FP,Week 186,n=39,46,16 | -9.4 (19.34) | -7.7 (26.69) | 3.5 (24.59)
  BI,Week 07,n=47,45,16: number analyzed (Participants) | 47 | 45 | 16
  BI,Week 07,n=47,45,16 | 2.8 (22.87) | 9.6 (28.09) | 4.2 (43.67)
  BI,Week 13,n=28,28,15: number analyzed (Participants) | 28 | 28 | 15
  BI,Week 13,n=28,28,15 | 6.0 (25.75) | 6.0 (35.20) | -4.4 (37.52)
  BI,Week 19,n=18,25,10: number analyzed (Participants) | 18 | 25 | 10
  BI,Week 19,n=18,25,10 | 5.6 (23.57) | 8.0 (25.96) | -3.3 (42.89)
  BI,Week 25,n=19,23,7: number analyzed (Participants) | 19 | 23 | 7
  BI,Week 25,n=19,23,7 | 7.0 (23.78) | 15.9 (31.57) | 9.5 (53.45)
  BI,Week 31,n=14,18,7: number analyzed (Participants) | 14 | 18 | 7
  BI,Week 31,n=14,18,7 | 2.4 (20.52) | 14.8 (30.73) | 9.5 (56.81)
  BI,Week 37,n=14,13,5: number analyzed (Participants) | 14 | 13 | 5
  BI,Week 37,n=14,13,5 | 9.5 (27.51) | 25.6 (30.89) | 26.7 (54.77)
  BI,Week 43,n=15,13,4: number analyzed (Participants) | 15 | 13 | 4
  BI,Week 43,n=15,13,4 | 4.4 (24.77) | 28.2 (38.12) | 8.3 (16.67)
  BI,Week 61,n=11,11,3: number analyzed (Participants) | 11 | 11 | 3
  BI,Week 61,n=11,11,3 | 6.1 (25.03) | 12.1 (26.97) | 33.3 (57.74)
  BI,Week 79,n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  BI,Week 79,n=3,2,2 | 0.0 (0.00) | 0.0 (0.00) | 33.3 (94.28)
  BI,Week 97,n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  BI,Week 97,n=4,5,3 | 8.3 (31.91) | 6.7 (27.89) | 44.4 (69.39)
  BI,Week 115,n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  BI,Week 115,n=2,6,3 | -16.7 (70.71) | 5.6 (25.09) | 55.6 (50.92)
  BI,Week 133,n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  BI,Week 133,n=2,1,2 | 16.7 (23.57) | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. | 83.3 (23.57)
  BI,Week 151,n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  BI,Week 151,n=0,2,0 |  | 16.7 (23.57) |
  BI,Week 169,n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  BI,Week 169,n=0,1,0 |  | 0.0 (NA) — NA indicates SD could not be calculated for a single participant. |
  BI,Week 186,n=39,46,16: number analyzed (Participants) | 39 | 46 | 16
  BI,Week 186,n=39,46,16 | -4.3 (30.76) | -0.7 (35.48) | 10.4 (41.67)
  DS,Week 07,n=47,45,16: number analyzed (Participants) | 47 | 45 | 16
  DS,Week 07,n=47,45,16 | -1.8 (19.73) | -1.0 (17.78) | -2.8 (12.17)
  DS,Week 13,n=28,28,15: number analyzed (Participants) | 28 | 28 | 15
  DS,Week 13,n=28,28,15 | -1.0 (16.22) | -3.2 (22.95) | 1.1 (25.65)
  DS,Week 19,n=18,25,10: number analyzed (Participants) | 18 | 25 | 10
  DS,Week 19,n=18,25,10 | 0.9 (14.91) | -6.4 (17.98) | -1.7 (20.63)
  DS,Week 25,n=19,23,7: number analyzed (Participants) | 19 | 23 | 7
  DS,Week 25,n=19,23,7 | -0.0 (16.25) | -3.6 (17.78) | -1.6 (25.20)
  DS,Week 31,n=14,18,7: number analyzed (Participants) | 14 | 18 | 7
  DS,Week 31,n=14,18,7 | -3.6 (10.59) | -10.5 (19.23) | -4.8 (23.88)
  DS,Week 37,n=14,13,5: number analyzed (Participants) | 14 | 13 | 5
  DS,Week 37,n=14,13,5 | -6.0 (12.22) | -9.8 (22.92) | -14.4 (16.01)
  DS,Week 43,n=15,13,4: number analyzed (Participants) | 15 | 13 | 4
  DS,Week 43,n=15,13,4 | -5.9 (12.51) | -14.5 (24.06) | -8.3 (26.64)
  DS,Week 61,n=11,11,3: number analyzed (Participants) | 11 | 11 | 3
  DS,Week 61,n=11,11,3 | -11.6 (12.29) | -7.6 (10.02) | -11.1 (16.67)
  DS,Week 79,n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  DS,Week 79,n=3,2,2 | -16.7 (11.11) | -2.8 (3.93) | -2.8 (27.50)
  DS,Week 97,n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  DS,Week 97,n=4,5,3 | -12.5 (15.30) | -3.3 (15.52) | -7.4 (25.05)
  DS,Week 115,n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  DS,Week 115,n=2,6,3 | -19.4 (3.93) | -7.4 (10.92) | -10.0 (16.59)
  DS,Week 133,n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  DS,Week 133,n=2,1,2 | -13.9 (11.79) | -5.6 (NA) — NA indicates SD could not be calculated for a single participant. | 8.3 (51.07)
  DS,Week 151,n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  DS,Week 151,n=0,2,0 |  | 5.6 (15.71) |
  DS,Week 169,n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  DS,Week 169,n=0,1,0 |  | -5.6 (NA) — NA indicates SD could not be calculated for a single participant. |
  DS,Week 186, n=39,46,16: number analyzed (Participants) | 39 | 46 | 16
  DS,Week 186, n=39,46,16 | -0.6 (17.28) | 2.5 (18.36) | 4.9 (24.50)
  SET,Week 07,n=47,45,16: number analyzed (Participants) | 47 | 45 | 16
  SET,Week 07,n=47,45,16 | 1.5 (9.21) | 0.4 (13.33) | 0.2 (15.49)
  SET,Week 13,n=28,28,15: number analyzed (Participants) | 28 | 28 | 15
  SET,Week 13,n=28,28,15 | 2.0 (10.44) | -1.7 (11.96) | 6.8 (23.69)
  SET,Week 19,n=18,25,10: number analyzed (Participants) | 18 | 25 | 10
  SET,Week 19,n=18,25,10 | 0.0 (10.40) | -1.2 (10.87) | 0.9 (9.04)
  SET,Week 25,n=19,23,7: number analyzed (Participants) | 19 | 23 | 7
  SET,Week 25,n=19,23,7 | 3.4 (8.41) | 0.1 (13.10) | 0.4 (6.45)
  SET,Week 31,n=14,18,7: number analyzed (Participants) | 14 | 18 | 7
  SET,Week 31,n=14,18,7 | 2.0 (6.07) | -2.9 (13.87) | 5.5 (11.12)
  SET,Week 37,n=14,13,5: number analyzed (Participants) | 14 | 13 | 5
  SET,Week 37,n=14,13,5 | 2.2 (6.91) | -6.0 (17.82) | -1.8 (4.04)
  SET,Week 43,n=15,13,4: number analyzed (Participants) | 15 | 13 | 4
  SET,Week 43,n=15,13,4 | 1.0 (8.81) | -5.6 (19.05) | -4.9 (5.76)
  SET,Week 61,n=11,11,3: number analyzed (Participants) | 11 | 11 | 3
  SET,Week 61,n=11,11,3 | -2.1 (12.32) | 1.9 (12.82) | 2.0 (9.84)
  SET,Week 79,n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  SET,Week 79,n=3,2,2 | 5.9 (11.40) | 9.1 (12.83) | -1.3 (4.45)
  SET,Week 97,n=4,5,3: number analyzed (Participants) | 4 | 5 | 3
  SET,Week 97,n=4,5,3 | -0.2 (5.42) | 5.0 (13.80) | -4.7 (3.44)
  SET,Week 115,n=2,6,3: number analyzed (Participants) | 2 | 6 | 3
  SET,Week 115,n=2,6,3 | 5.7 (13.36) | 0.7 (7.21) | -1.0 (7.09)
  SET,Week 133,n=2,1,2: number analyzed (Participants) | 2 | 1 | 2
  SET,Week 133,n=2,1,2 | 5.7 (13.36) | -7.4 (NA) — NA indicates SD could not be calculated for a single participant. | -8.1 (5.24)
  SET,Week 151,n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  SET,Week 151,n=0,2,0 |  | 0.0 (15.71) |
  SET,Week 169,n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  SET,Week 169,n=0,1,0 |  | -11.1 (NA) — NA indicates SD could not be calculated for a single participant. |
  SET,Week 186,n=39,46,16: number analyzed (Participants) | 39 | 46 | 16
  SET,Week 186,n=39,46,16 | 4.0 (10.98) | 4.0 (12.61) | 3.7 (10.75)

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious adverse events (SAEs) and (>=5%) non-serious AEs (Non-SAEs) were collected from the start of study treatment until maximum of 186 weeks for main study and up to approximately 325 weeks for PACT phase.
Description: SAEs & non-SAEs for Full Safety Population comprised all participants who received atleast 1 dose of treatment.3 out of 221 participants didn't receive treatment & thus excluded from reporting. All-cause mortality for Full Safety Population comprised all randomized participants whether or not randomized treatment was administered.
Arm/Group | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized) | PACT Phase: GSK2857916 2.5 mg/kg (Frozen Liquid) | PACT Phase: GSK2857916 3.4 mg/kg (Frozen Liquid)
All-Cause Mortality (participants affected / at risk) | 70/97 | 80/99 | 16/25 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 43/95 | 53/99 | 15/24 | 1/1 | 2/2
Other Adverse Events (participants affected / at risk) | 93/95 | 96/99 | 24/24 | 0/1 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) (N=95) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) (N=99) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized) (N=24) | PACT Phase: GSK2857916 2.5 mg/kg (Frozen Liquid) (N=1) | PACT Phase: GSK2857916 3.4 mg/kg (Frozen Liquid) (N=2)
Pneumonia (Infections and infestations) | 7 (8) | 14 (16) | 1 (1) | 0 | 0
Pyrexia (General disorders) | 7 (8) | 5 (7) | 0 (0) | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 3 (3) | 3 (3) | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 1 (1) | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (4) | 2 (2) | 0 (0) | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 | 0
Sepsis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 | 0
Cellulitis (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 | 0
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 | 0
General physical health deterioration (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 | 0
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 | 0
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 | 0
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 | 0
Vascular device infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Brain abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Gastric fibrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Herpes simplex pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Infective keratitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Keratopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nocardiosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study: GSK2857916 2.5 mg/kg (Frozen Liquid) (N=95) | Main Study: GSK2857916 3.4 mg/kg (Frozen Liquid) (N=99) | Main Study: GSK2857916 3.4 mg/kg (Lyophilized) (N=24) | PACT Phase: GSK2857916 2.5 mg/kg (Frozen Liquid) (N=1) | PACT Phase: GSK2857916 3.4 mg/kg (Frozen Liquid) (N=2)
Keratopathy (Eye disorders) | 67 (267) | 74 (320) | 23 (100) | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (34) | 44 (73) | 8 (12) | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 25 (28) | 36 (49) | 8 (14) | 0 | 0 (0)
Vision blurred (Eye disorders) | 22 (37) | 30 (50) | 8 (13) | 0 | 0
Nausea (Gastrointestinal disorders) | 24 (29) | 32 (40) | 2 (3) | 0 | 0
Fatigue (General disorders) | 15 (19) | 28 (37) | 12 (13) | 0 | 0
Aspartate aminotransferase increased (Investigations) | 21 (26) | 24 (30) | 6 (8) | 0 | 0
Pyrexia (General disorders) | 18 (21) | 22 (29) | 4 (6) | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (24) | 16 (19) | 4 (6) | 0 | 0
Dry eye (Eye disorders) | 14 (18) | 19 (21) | 5 (10) | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 12 (16) | 19 (21) | 5 (5) | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 10 (12) | 20 (24) | 4 (4) | 0 | 0
Headache (Nervous system disorders) | 11 (12) | 17 (22) | 5 (6) | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 19 (20) | 3 (4) | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 12 (12) | 6 (6) | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 11 (14) | 15 (15) | 4 (4) | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 10 (11) | 15 (17) | 4 (5) | 0 | 0
Platelet count decreased (Investigations) | 15 (18) | 11 (26) | 3 (3) | 0 | 0
Vomiting (Gastrointestinal disorders) | 8 (11) | 21 (23) | 0 (0) | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 17 (21) | 1 (1) | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 10 (10) | 14 (14) | 2 (2) | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 15 (16) | 9 (10) | 2 (2) | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 7 (17) | 18 (27) | 1 (4) | 0 | 0
Constipation (Gastrointestinal disorders) | 12 (13) | 9 (9) | 4 (5) | 0 | 0
Lymphocyte count decreased (Investigations) | 13 (15) | 10 (13) | 2 (3) | 0 | 0
Blood creatinine increased (Investigations) | 10 (11) | 11 (14) | 2 (2) | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 9 (10) | 11 (11) | 1 (1) | 0 | 0
Hypertension (Vascular disorders) | 9 (10) | 10 (11) | 2 (6) | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 (6) | 12 (14) | 4 (4) | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8) | 12 (16) | 1 (1) | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 12 (13) | 3 (7) | 0 | 0
Neutrophil count decreased (Investigations) | 7 (10) | 11 (13) | 2 (2) | 0 | 0
Intraocular pressure increased (Investigations) | 6 (10) | 8 (8) | 5 (6) | 0 | 0
Photophobia (Eye disorders) | 7 (12) | 9 (16) | 3 (3) | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 7 (10) | 8 (11) | 3 (3) | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (7) | 3 (3) | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 9 (23) | 7 (7) | 1 (1) | 0 | 0
Asthenia (General disorders) | 3 (3) | 11 (11) | 2 (2) | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 9 (9) | 7 (8) | 0 (0) | 0 | 0
Urinary tract infection (Infections and infestations) | 6 (7) | 9 (16) | 1 (1) | 0 | 0
White blood cell count decreased (Investigations) | 7 (8) | 9 (11) | 0 (0) | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 4 (5) | 7 (8) | 4 (4) | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (9) | 7 (11) | 3 (4) | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (9) | 1 (1) | 0 | 0
Chills (General disorders) | 8 (8) | 4 (4) | 2 (2) | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 9 (10) | 0 (0) | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 8 (12) | 1 (1) | 0 | 0
Visual acuity reduced (Eye disorders) | 5 (8) | 5 (5) | 3 (3) | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (7) | 6 (8) | 1 (1) | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 6 (6) | 5 (5) | 1 (1) | 0 | 0
Oedema peripheral (General disorders) | 5 (5) | 4 (10) | 3 (5) | 0 | 0
Proteinuria (Renal and urinary disorders) | 5 (11) | 3 (21) | 3 (3) | 0 | 0
Weight decreased (Investigations) | 8 (8) | 2 (2) | 1 (1) | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 (6) | 4 (5) | 0 (0) | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 8 (8) | 2 (2) | 0 | 0
Urine albumin/creatinine ratio increased (Investigations) | 2 (2) | 8 (8) | 0 (0) | 0 | 0
C-reactive protein increased (Investigations) | 3 (3) | 5 (5) | 1 (1) | 0 | 0
Dizziness (Nervous system disorders) | 1 (1) | 7 (8) | 1 (1) | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 2 (2) | 0 | 0
Insomnia (Psychiatric disorders) | 6 (6) | 1 (1) | 2 (2) | 0 | 0
Pain (General disorders) | 5 (5) | 4 (4) | 0 (0) | 0 | 0
Pneumonia (Infections and infestations) | 2 (2) | 5 (5) | 2 (2) | 0 | 0
Blepharitis (Eye disorders) | 2 (3) | 6 (6) | 0 (0) | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 5 (13) | 3 (3) | 0 (0) | 0 | 0
Bronchitis (Infections and infestations) | 6 (6) | 2 (2) | 0 (0) | 0 | 0
Diplopia (Eye disorders) | 2 (3) | 4 (5) | 2 (2) | 0 | 0
Eye pruritus (Eye disorders) | 2 (2) | 5 (10) | 1 (1) | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 0 (0) | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 2 (2) | 0 | 0
Chest pain (General disorders) | 2 (2) | 2 (2) | 3 (3) | 0 | 0
Depression (Psychiatric disorders) | 5 (5) | 2 (3) | 0 (0) | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 2 (2) | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 1 (1) | 0 | 0
Confusional state (Psychiatric disorders) | 0 (0) | 5 (6) | 1 (1) | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 (1) | 5 (6) | 0 (0) | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 2 (2) | 0 | 0
Haematuria (Renal and urinary disorders) | 2 (8) | 1 (1) | 2 (2) | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2) | 0 | 0
Blood bilirubin increased (Investigations) | 1 (1) | 1 (2) | 2 (2) | 0 | 0
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03525678/Prot_004.pdf
  • Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03525678/SAP_003.pdf